Trial: SAP Version: 1.1

STRIVE

Version Date: 03/08/2022



# STATISTICAL ANALYSIS PLAN

Effectiveness and cost of integrating a protocol with use of Liraglutide 3.0mg into an obesity service (STRIVE Study)

**SAP Version:** 

1.1

Date:

03/08/2022

Based on protocol: Effectiveness and cost of integrating a protocol with use of Liraglutide 3.0mg into an obesity service, Version 7.0; 29/01/2021

**Sponsor Reference No:** 

**UNOLE 0626** 

**Ethics Ref:** 

17 NW 0517

**EudraCT Number:** 

2017-002998-20

Universal Trial Number (UTN):

U1111-1189-5726

**Sponsor:** 

Name: University of Leicester

Address: University Road, Leicester, LE1 7RH

**SAP Author:** 

Name: Dr Danielle Bodicoat

Organisation: Independent researcher

**Trial Statistician:** 

Name: Dr Shaun Barber

Organisation: Leicester Clinical Trials Unit, University of Leicester

**Chief Investigator:** 

Name: Professor Melanie Davies

Organisation: Diabetes Research Centre, University of Leicester

Trial Manager:

Name: Sarah Clarke

Organisation: Leicester Diabetes Centre, University Hospitals of

Leicester NHS Trust

Trial:

STRIVE

SAP Version: 1.1 Version Date: 03/08/2022



# **Revision History**

| Version | Date | Author(s) and Role | Summary of Changes/Comments |
|---|---|---|---|
| 0.1 | 02/11/2017 | Shaun Barber | Started drafting SAP |
| 0.2 | 13/02/2022 | Danielle Bodicoat | Completion of draft SAP ready for finalisation |
| 0.3 | 08/03/2022 | Danielle Bodicoat | Update of draft SAP based on initial review |
| 0.4 | 01/04/2022 | Danielle Bodicoat | Update of draft SAP based on review |
| 0.5 | 05/07/2022 | Shaun Barber | Update of draft SAP based on review |
| 1.0 | 12/07/2022 | Shaun Barber | Updated and finalised draft as v1.0 based on review |
| 1.1 | 01/08/2022 | Shaun Barber | Updated the definition of Glycaemic Status at baseline and follow-up add more detail in terms of medication and previous history of diabetes or pre-diabetes. Addition of summarising Glycaemic Status at follow-up by baseline status. Addition of summarising the proportion that met diabetes HbA1c targets (<6.5% and <7.0%) |



# SAP approval for finalised version:

| Trial Statistician | Shaun Barber | |
|---------------------|----------------|------------|
| | Chan Bobs. | 03/08/2022 |
| | Signature | Date |
| Chief Investigator | Melanie Davies | |
| | 161 | 12/10/2022 |
| | Signature | Date |
| Senior Statistician | Cassey Brookes | |
| | Rookey | |
| | | 03/08/2022 |
| | Signature | Date |




#### LIST OF ABBREVIATIONS

ADA American Diabetes Association

AE Adverse Event
BMI Body Mass Index
CSR Clinical Study Report

EQ-5D European Quality of Life -5 Dimensions

GP General Practitioner

HSRUQ Health Services and Resources Use Questionnaire

ICH International Conference on Harmonization of Technical Requirements for

Registration of Pharmaceuticals for Human Use

IFG Impaired fasting glycaemia IGT Impaired glucose tolerance

IPAQ-Long International Physical Activity Questionnaire-Long

ITT Intention-to-treat

IWQOL-Lite Impact of Weight on Quality of Life-Lite

LIRA Liraglutide

OSA Obstructive Sleep Apnoea
PHQ-9 Patient Health Questionnaire-9

SAE Serious Adverse Event SAP Statistical Analysis Plan

TSQM Treatment Satisfaction Questionnaire for Medication

TZD Thiazolidinediones






#### Contents

| 1 | Introd | uction | 8 |
|---|---------|--------------------------------------------------|----------|
| | 1.1 Stu | dy Objectives | 8 |
| | 1.1.1 | Primary Aim | 9 |
| | 1.1.2 | Primary Objectives | 8 |
| | 1.1.3 | Secondary Objectives | 9 |
| | 1.1.4 | Subgroup Objectives | 9 |
| | 1.2 Stu | dy Design | 9 |
| | 1.2.1 | Overview | 9 |
| | 1.2.2 | Participants | 12 |
| | 1.2.3 | Treatment groups | 12 |
| | 1.2.4 | Sample size | 14 |
| | 1.2.5 | Randomisation and blinding | 15 |
| | 1.3 Vis | it schedule | 15 |
| 2 | Outcor | nes and other variables | _16 |
| _ | | mary Endpoint | |
| | 2.1.1 | Definition and Derivation of Primary Endpoint | |
| | 2.1.2 | Hypothesis to be investigated | |
| | | condary Endpoints | |
| | 2.2.1 | Definition and Derivation of Secondary Endpoints | |
| | | ogroups and/or interactions | |
| | | mpliance | |
| | | ner | |
| 3 | Analyz | sis Sets/Populations | 25 |
| 3 | 3.1 Dis | sposition of participants | 23<br>25 |
| | | tocol deviations | |
| | | oulations | |
| | 3.3.1 | Complete Cases Population | |
| | 3.3.2 | Intention-To-Treat Population | |
| | 3.3.3 | Per Protocol Population | |
| | 3.3.4 | Responder Population | |
| | 3.3.5 | Safety Population | |
| _ | | • • | |
| 4 | | al Issues for Statistical Analysis | |
| | | alysis Groups | |
| | | ssing Data | |
| | | rived/ Computed Variables | |
| | | ltiple Testing | |
| | | alysis Software | |
| | | tistical Significance | |
| | | tliers | |
| 5 | | ical Methodology | |
| | | sposition | |
| | | erim analysis | |
| | | mographic and Baseline Characteristics | |
| | | mary Outcome Analysis | |
| | 5.4.1 | Primary Analysis of Primary Outcome | 31 |




| 5.4.2 | Secondary Analyses of Primary Outcome | 31 |
|---|---|---|
| 5.4.3 | Sensitivity Analyses | 31 |
| 5.4.4 | | |
| 5.5 | Secondary Outcome Analyses | |
| 5.5.1 | | |
| 5.5.2 | | 32 |
| 5.5.3 | Subgroup AnalysesSubgroup Analyses | |
| 5.6<br>5.7 | Figures to be produced | 33 |
| 5.8 | Changes to the Planned Analysis | 33 |
| | ty and Adverse events (AEs) | |
| 7 Refe | erences | 36 |
| 8 App | endix 1: Scoring for King's College Obesity Staging System | 37 |
| 9 App | endix 2: Scoring for PHQ-9 Questionnaire | 38 |
| 10 A | ppendix 3: Scoring for Epworth Sleepiness Scale | 39 |
| 11 A | ppendix 4: Scoring for Stop Bang Questionnaire | 40 |
| 12 A | ppendix 5: Definitions of hypoglycaemia | 41 |
| 13 A | ppendix 6: IPAQ scoring system | 43 |
| 14 A | ppendix 7 Definitions for adherence of participants with the LIRA 3m | ıg45 |
| 14.1 | 52 weeks | 45 |
| 14.2 | 104 weeks | 46 |
| 15 A | ppendix 8: Baseline and follow-up Glycaemic Status Definitions | 47 |
| 15.1 | Baseline Glycaemic Status | 47 |
| 15.2 | Follow-up Glycaemic Status | |
| 16 A | ppendix 9: Templates for Tables | 49 |
| 16.1 | Disposition | 49 |
| 16.2 | Protocol deviations | 49<br>50 |
| 16.3 | Summary of continuous baseline characteristics | |
| 16.4<br>16.5 | Summary of categorical baseline characteristics | 52 |
| withou | at primary outcome data | 54 |
| 16.6 | Comparison of categorical baseline characteristics between those with and | |
| | t primary outcome data | 56 |
| 16.7 | Analysis of primary outcome | 58 |
| 16.8 | Analysis of secondary categorical anthropometric outcomes | 59 |
| 16.9 | Analysis of secondary continuous anthropometric outcomes | 61 |
| 16.10 | Summary of other categorical secondary outcomes | 66<br>حم |
| 16.11 | Summary of other secondary continuous outcomes | ۷۵<br>7۵ |
| 16.12 | Summary of categorical safety outcomes | <i>ነ 9</i><br>የበ |
| 16.13<br>16.14 | Summary of continuous safety outcomes | 83 |
| | Summary of categorical compliance outcomes | (7.7 |
| 16.15 | Summary of categorical compliance outcomes | 85 |

Trial:

STRIVE

SAP Version: 1.1







#### 1 Introduction

This Statistical Analysis Plan (SAP) describes the planned analysis and reporting for the following study: Effectiveness and cost of integrating a protocol with use of Liraglutide 3.0mg into an obesity service (STRIVE Study). The structure and content of this SAP provides sufficient detail to meet the requirements identified by the FDA and International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH): Guidance on Statistical Principles in Clinical Trials. All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association and the Royal Statistical Society for statistical practice.

The reader of this SAP is encouraged also to read the clinical trial protocol.

The purpose of this SAP is to outline the planned analyses that are to be performed on the data to support the completion of the Clinical Study Report (CSR), i.e., this SAP only covers the final analyses. The SAP will be amended if there are substantial changes to the planned analyses, and in any case will be finalized and signed off before the database lock for this study.

Exploratory post-hoc or unplanned analyses not necessarily identified in this SAP may be performed on these data as required. These analyses will be clearly identified in the CSR and in any subsequent publications of the data that include post-hoc or unplanned analyses.

It is planned that health economics analyses will be performed. These will be handled separately and are not described in this SAP.

Interim analyses have not been performed for this study. Safety analyses were conducted for the Data Monitoring Committee reports, but no efficacy analyses took place.

Throughout the document, any verbatim text from the protocol is provided inside a box, i.e.:

Text from the protocol

# 1.1 Study Objectives

#### 1.1.1 Primary Objectives

The primary objective will be to compare the proportion of participants with severe and complicated obesity (defined as  $BMI \ge 35 \text{ kg/m}^2$  with at least one major obesity-related comorbidity) achieving weight loss  $\ge 15\%$  at 1 year (52 weeks) with a targeted prescribing pathway (i.e. use of LIRA 3mg according to a pre-specified protocol in combination with standard care provided in Tier 3 services) versus standard care provided in Tier 3 services alone.

Trial:

**STRIVE** 

SAP Version: 1.1




#### 1.1.2 Primary Aim

The aim of the study is to compare the effectiveness, budget impact, and cost-effectiveness between two treatment pathways (standard care vs a targeted prescribing pathway plus standard care) in a real-world setting among otherwise largely unselected patients.

The secondary objectives are to compare the targeted prescribing pathway and standard care in terms of:

- 1. improving obesity-related co-morbidities (obstructive sleep apnoea, prediabetes, diabetes, hypertension, dyslipidaemia, depression)
- 2. referral rates to other obesity interventions
- 3. long-term maintenance (defined as the proportion of participants maintaining weight loss of ≥15% at 104 weeks among those who achieved ≥15% weight loss at 52 weeks)
- 4. budget impact on a Tier 3 weight management service
- 5. long-term cost-effectiveness
- 6. direct healthcare costs in terms of admissions, frequency, and cost of appointments
- 7. safety-related outcomes
- 8. adherence
- 9. patient satisfaction.

#### 1.1.3 Secondary Objectives

Secondary objectives number 4-6 will be dealt with as part of the health economics analysis and are not included in this SAP.

#### 1.1.4 Subgroup Objectives

None

## 1.2 Study Design

#### 1.2.1 Overview

A 26 month, parallel, two group, open-label, real-world, randomized controlled trial design for patients with severe and complex obesity who are referred to a Tier 3 obesity service (including patients who are referred to a Tier 3 service as part of the bariatric surgery pathway). The total duration of participation will be 104 weeks (+/-2 weeks). Figure 1 shows an overview of the study design.

The first 52 weeks of the study (after randomisation) will determine whether using the




targeted prescribing pathway in a Tier 3 setting will result in more participants attaining ≥15% weight loss compared with standard care. The purpose of the long-term (52-104 weeks) follow-up is to examine whether LIRA 3mg will help the "early and good" responders to maintain weight loss ≥15% in comparison with the control group over a longer period of time compared with standard care. Further, budget impact, cost-effectiveness, improvement in obesity-related co-morbidities, complementary aspects of safety, effectiveness, adherence, and treatment satisfaction of both treatment groups will be assessed and compared.

Participants will be randomised in a 2:1 fashion (2 intervention: 1 control) to either 1) the intervention of targeted prescribing pathway (obesity-specialist care plus targeted use of Liraglutide 3.0mg [LIRA 3mg] with pre-specified stopping rules for the medication) plus standard care, or 2) control (standard care). All participants will be analysed in the group to which they are randomised; in particular, participants in the intervention group who stop receiving LIRA 3mg will remain in the intervention group and will continue to receive standard care for the remainder of the study as per the targeted prescribing pathway (albeit, the part of the pathway where LIRA 3mg is not prescribed; see Figure 1).

The study is intentionally designed to reflect a pragmatic "real-world" scenario and each Tier 3 provider may require a different number of visits for their programme. However, study appointments for data collection, titration reviews, application of the stopping rules of LIRA 3mg, and dispensing were standardised for all of the five sites. Where participants were lost to follow up or missed a study visit, the study team attempted to access data for weight measurements from existing hospital, GP or health records, where appropriate consent was in place, to ensure that the primary outcome was as complete as possible.





#### 1.2.2 Participants

#### **Inclusion Criteria**

To be considered eligible to participate in this study, a patient must:

- be aged between 18-75 years old (inclusive)
- understand written and spoken English
- be able to give informed consent
- have a BMI ≥35 kg/m<sup>2</sup>
- have been referred to the Tier 3 service in one of the participating sites
- have a stable body weight (less than 5kg self-reported change during the previous 12 weeks)
- have at least one of prediabetes, diabetes, hypertension, and/or obstructive sleep apnoea, as defined below:
  - prediabetes (defined as established diagnosis of impaired fasting glycaemia (IFG) from GP and/or established diagnosis of impaired glucose tolerance (IGT) from GP and/or HbA1C 42-47 mmol/mol (6-6.4%) without glucose lowering medications, at a blood test during the last 6 months)
  - diabetes (defined as established diagnosis of Type 2 diabetes from GP and/or HbA1C ≥48 mmol/mol (≥6.5%) at a blood test during the last 6 months] and/or being treated with any combination of lifestyle, metformin, sulphonylureas, Thiazolidinediones (TZDs) or SGLT-2)
  - hypertension treated (defined as being on antihypertensive treatment with or without a diagnosis of hypertension from GP) or untreated (defined as Systolic Blood Pressure ≥140 mmHg at two consecutive visits at the Tier 3 clinic),
  - obstructive sleep apnoea (on CPAP or established diagnosis of Apnoea
     Hypopnoea Index ≥15 at sleep studies during the last 12 months).

Exclusion criteria are stated in the protocol, and cover contradictions to LIRA 3mg and criterion that would be likely to prevent full participation in the study protocol.

#### 1.2.3 Treatment groups

#### 1.2.3.1 Intervention group (Targeted Prescribing Pathway)

The NHS Weight Management pathway is divided into four distinct tiers:

**Tier 1:** health promotion

**Tier 2:** lifestyle interventions

Tier 3: specialist multidisciplinary weight management services



#### **Tier 4:** bariatric surgery

Across the UK, each region has a specialist Tier 3 obesity and/or weight management service or equivalent, usually referred to as Tier 3. This includes a clinician led multidisciplinary team approach, potentially including a specialist physician, nurse, dietician, psychologist, physiotherapist, etc. From this point forwards, Tier 3 specialist weight management and/or equivalent services will be referred to as 'Tier 3' throughout the remainder of this protocol.

Participants in the intervention group will receive the same standard care as those in the control group, i.e. the best medical practice delivered by the Tier 3 service at each site.

Additionally, at baseline, LIRA 3mg will be prescribed to all of the participants in the intervention group at a starting dose of 0.6mg daily. Dose escalation of Liraglutide will occur according to a pre-specified titration protocol, from 0.6mg to a maximum of 3.0mg daily. Liraglutide dose will be initiated at 0.6mg and then increased to 1.2mg in Week 2, 1.8mg in Week 3, 2.4mg in Week 4, and 3.0mg in Week 5. Participants in the intervention group will be aware that the LIRA 3mg treatment may be stopped at various time points throughout the duration of the study and that continued use of LIRA 3mg is based upon their response to the treatment in terms of them achieving pre-defined weight loss targets at 16, 32 and 52 weeks. Specifically, participants in the intervention group will continue to be prescribed LIRA 3mg for the 104 week duration of the study, unless one of the following stopping rules applies:

#### 1<sup>st</sup> stopping rule

After 16 weeks (± 14 days) on the medication, only those participants who have lost ≥5% of their baseline weight will be offered further treatment with LIRA 3mg for another 16 weeks. Participants who have not met this weight loss target will have their LIRA 3mg treatment stopped but will still continue in the targeted prescribing pathway but will receive standard care only during the remainder of the study.

#### 2<sup>nd</sup> stopping rule

After 32 weeks (± 14 days) on the medication, only those participants who have lost ≥10% of their baseline weight and are still on treatment with LIRA 3mg will be offered another 20 weeks on LIRA 3mg. Participants who have not met this weight loss target will have their LIRA 3mg treatment stopped but will still continue in the targeted prescribing pathway but will receive standard care only during the remainder of the study.

# 3<sup>rd</sup> stopping rule

After the first year of treatment (week 52; ± 14 days), only those participants who have lost ≥15% of their baseline weight and are still on treatment with LIRA 3mg will be offered another 52 weeks on LIRA 3mg. Participants who have not met this weight loss target will



have their LIRA 3mg treatment stopped and will still continue in the targeted prescribing pathway but will receive standard care only during the remainder of the study.

Participants who fail to reach the pre-defined weight-loss targets to continue LIRA 3mg treatment, or who choose to stop receiving LIRA 3mg, will continue to be offered the standard care provided by the Tier 3 service. These participants will still attend the Clinical Review Visits but not the additional visits for participants who are still on LIRA 3mg (e.g. Weeks 65 & 91) because these visits will not be relevant to them; visits at Weeks 65 and 91 are intended to provide a new prescription of LIRA 3mg and to discuss adherence and any side effects).

Participants will remain routinely in the Tier 3 service in-line with NICE guidance throughout the duration of the research study. Participants may be offered treatment options within the duration of the study, including bariatric surgery, as per NICE guidance and according to the decision of the local Tier 3 Multidisciplinary Team.

#### 1.2.3.2 Control group (standard care)

Participants in the control group will follow the best medical care provided by the Tier 3 service at the relevant site. This typically involves dietary advice to reduce energy intake (and may include a period of partial or total meal replacement), accompanied – if available – by a physical activity programme, both supported by behavioural change techniques with regular professional contacts. The nature of the standard care will vary between the different Tier 3 services at each site, as this is a pragmatic 'real-world' study. Clinician input will include the medical assessment of participants for severe and complicated obesity and the prescription of anti-obesity drugs (such as Orlistat) as per local Tier 3 service policy. As with the LIRA 3mg group those patients taking antihypertensive or antidepressant medication will be assessed and it will be at the clinician's discretion as to whether these medications are changed. Participants will remain routinely in the Tier 3 service in line with NICE guidance throughout the duration of the research study. Participants may be offered treatment options within the duration of the study, including bariatric surgery, as per NICE guidance and according to the decision of the local Tier 3 Multidisciplinary Team.

#### 1.2.4 Sample size

Based on previous studies, it is expected that at one year approximately 5% of the participants in the standard care group will have achieved ≥15% weight loss (likely range: 3%-5%). An achievable target for ≥15% weight loss at one year in the intervention group is 16% (likely range: 14%-20%). Based on these proportions, 25% drop out, 5% alpha and a 2:1 randomisation ratio with the higher proportion of participants being randomised to the



intervention group, we would need to recruit 392 participants (261 intervention group; 131 standard care) to have 80% power to detect a significant difference between the groups at one year. With 261 participants randomised to the intervention group, and based on 16% achieving ≥15% weight loss at 12 months, an estimated 40 participants in the intervention group will be eligible for the responder analyses. All 131 participants in the standard care group will be eligible for the responder analyses.

#### 1.2.5 Randomisation and blinding

This is an open-label study and so there is no blinding.

Randomisation will be conducted through a validated online system (sealedenvelope.com) provided through the LCTU. Eligible participants will be randomly assigned at their Baseline Visit (Day 0) in a 2:1 ratio to participate in a Tier 3 service with:

1) Targeted prescribing pathway - The use of once daily subcutaneous injections of Liraglutide (if they meet the pre-specified criteria), starting at a dose of 0.6 mg with gradual and pre-specified increments to 3.0mg

or

2) Control Group - No additional treatment.

A 2:1 ratio will be used so that a sufficient number of responders will be available for responder analyses. Randomisation will be stratified by centre and BMI ( $\geq$ 45kg/m<sup>2</sup>; <45kg/m<sup>2</sup>).

Participants will be informed of their randomisation assignment during the Baseline Visit. A letter will be sent to the participant's GP notifying them of their patient's participation in the study. Both the participant and their GP will have the randomisation assignment confirmed by letter.

#### 1.3 Visit schedule

The original visit schedule was as follows:

- Screening and Consent Visit (Day -42 to -1)
- Data Collection Visits All participants
  - Baseline Visit (Day 0) including randomization and treatment initiation for participants randomized to the intervention arm
  - Week 52
  - o Week 104

UNIVERSITY OF LEICESTER

Clinical Review (safety and retention) Visits – All participants

- Weeks 2, 4, 8, 12, 16, 20, 32, 40, and 78
- Additional Clinical Review (safety and retention) Visits for LIRA 3mg group
  - Weeks 65 and 91

In response to the COVID-19 global pandemic, an interim time point for the quality-of-life questionnaires was added. The following questionnaires were sent out to all participants during the COVID-19 pandemic:

- Health Services and Resources Use Questionnaire (HSRUQ)
- Treatment Satisfaction Questionnaire for Medication (TSQM)
- European Quality of Life -5 Dimensions (EQ-5D)
- Impact of Weight on Quality of Life-Lite (IWQOL-Lite)
- International Physical Activity Questionnaire-Long (IPAQ-Long)
- Patient Health Questionnaire-9 (PHQ-9).

Where possible, the week 52 visit continued to be scheduled within the  $\pm$  14 days study visit window, however to aid retention and to help maximise data collection for the study primary end point, the week 52 visit window could be extended to  $\pm$  3 months. Where it was not possible to conduct a week 52 visit (e.g., because of COVID-19 restrictions in place at the time), weight data were obtained from the participant's hospital, GP or health record instead where a measurement was available within a window of +/- 12 weeks from the scheduled week 52 visit to ensure that the primary outcome was as complete as possible.

#### 2 Outcomes and other variables

#### 2.1 Primary Endpoint

#### 2.1.1 Definition and Derivation of Primary Endpoint

Binary outcome indicating whether weight loss of ≥15% was achieved at 52 weeks.

Percentage weight loss at 52 weeks will be derived for each participant using the following formula:

$$\frac{(weight_{baseline\ visit}-weight_{52\ week\ visit})}{weight_{baseline\ visit}}\ x\ 100$$

The primary endpoint will then be coded as 1 if the percentage weight loss at 52 weeks is ≥15%, and as 0 otherwise.



As stated in section 1.3 where weight is not available from week 52 visit, weight from routinely collected data will be used instead if possible.

## 2.1.2 Hypothesis to be investigated

The primary hypothesis is that a targeted prescribing pathway using LIRA 3mg according to a pre-specified protocol in combination with standard care provided in Tier 3 services will be associated with more participants achieving weight loss of ≥15% at 1 year than receiving standard care provided in Tier 3 services alone.



# 2.2 Secondary Endpoints

# 2.2.1 Definition and Derivation of Secondary Endpoints

| https://www.qualityoflifeconsulting.com/iwqol-lite.html with change from baseline | · | (IWQOL-Lite) | |
|---|---|---|---|
| Transformed total score on scale of 0-100 scored as per | 52, 104 | Impact of Weight on Quality of Life-Lite | |
| Scored as per https://www.unmc.edu/centric/_documents/EQ-5D-5L.pdf with change from baseline value analysed | 52, 104 | Quality of life (EQ5D) – Visual Analogue Scale | |
| Scored as per https://www.unmc.edu/centric/_documents/EQ-5D-5L.pdf with change from baseline value analysed separately for each dimension | 52, 104 | Quality of life (EQ5D) – Descriptive System | |
| disease), 2 (established disease), 3 (advanced disease) with baseline values also presented | | System assessment | |
| Scored as per Staging System (Appendix 1) as Stage 0 (normal health), 1 (at risk of | 52, 104 | Score on King's College Obesity Staging | |
| | tments (General) | Obesity-related co-morbidities and their treatments (General) | |
| | | from baseline | |
| Follow-up waist circumference – baseline waist circumference | 52, 104 | Absolute change in waist circumference (cm) | |
| | | baseline | |
| Follow-up BMI – baseline BMI | 52, 104 | Absolute change in BMI (kg/m²) from | 1 |
| otherwise, only calculated for those who lost ≥15% of baseline weight at 52 weeks. | | those who lost ≥15% at 52 weeks | |
| Binary indicator of 1 if relative change in weight from baseline is ≥15% loss, 0 | 104 | Maintenance of weight loss of ≥15% among | |
| or ≥15%, respectively), 0 otherwise | | | _ |
| Binary indicator of 1 if relative change in weight from baseline is ≥5% loss (or ≥10% | 16, 32, 52, 104 | Weight loss of ≥5%, ≥10% and ≥15% | - |
| (Baseline weight – follow-up weight)/baseline weight * 100 | 16, 32, 52, 104 | Relative change in weight (%) from baseline | |
| Follow-up weight baseline weight | 16, 32, 52, 104 | Absolute change in weight (kg) from baseline | |
| | | Anthropometric endpoint | |
| s) Endpoint derivation | Time point (weeks) | Endpoint | |
| | | | 7 |



| definitions. | | |
|---|---|---|
| separately as well as for all individuals, see Appendix 8 for Glycaemic Status | | |
| Follow-up HbA1c – baseline HbA1c. Will be calculated for each Glycaemic Status | 52, 104 | Change in HbA1C from baseline (mmol/mol) |
| petes/Diabetes) | ments (Prediak | Obesity-related co-morbidities and their treatments (Prediabetes/Diabetes) |
| | | or for participants on fixed pressures CPAP |
| hour can be measured using PSG and is called the oxygen desaturation index (ODI).) | | with sleep apnoea who cannot tolerate CPAP |
| Recorded as integer in MACRO (The average number of desaturation episodes per | 52, 104 | Oxygen desaturation index for participants |
| on average, each nour.) | | for participants on fixed pressures CPAP |
| breathing) plus the number of hypopneas (periods of shallow breathing) occurring, | | sleep apnoea who cannot tolerate CPAP or |
| Recorded as an integer in MACRO (AHI = sum of the number of apneas (pauses in | 52, 104 | Apnoea Hypopnea Index for participants with |
| presented | | |
| Binary indicator of 1 if participant is on CPAP, 0 otherwise with baseline values also | 52, 104 | On CPAP |
| Total score generated as per Appendix 4 with change from baseline analysed | 52, 104 | Stop Bang questionnaire |
| baseline values also presented | | |
| Scored as per Appendix 4 as no OSA (0-2), possible OSA (3-4), likely OSA (5-8) with | 52, 104 | Stop Bang questionnaire |
| Total score generated as per Appendix 3 with change from baseline analysed | 52, 104 | Epworth Sleepiness Scale |
| values also presented | | |
| Scored as per Appendix 3 as binary outcome for possible OSA or not with baseline | 52, 104 | Epworth Sleepiness Scale |
| ctive Sleep Apnoea; OSA) | ments (Obstrue | Obesity-related co-morbidities and their treatments (Obstructive Sleep Apnoea; OSA) |
| Total score generated as per Appendix 2 with change from baseline analysed | 52, 104 | Patient Health Questionnaire-9 (PHQ-9) |
| also presented | | |
| depression, moderately severe depression, severe depression with baseline values | | |
| Scored as per Appendix 2 as minimal depression, mild depression, moderate | 52, 104 | Patient Health Questionnaire-9 (PHQ-9) |
| value analysed | | |



| Change in HbA1C from baseline (%) | 52. 104 | Follow-up HbA1c – baseline HbA1c Will be calculated for each baseline Glycaemic |
|---|---|---|
| | | Status separately as well as for all individuals, see Appendix 8 for Glycaemic Status |
| | | definitions) |
| Glycaemic Status | 52, 104 | Individuals are classified as having Diabetes remission, Diabetes, Pre-diabetes or |
| | | Normoglycaemia. The Glycaemic Statuses will be summarised overall as well as for |
| | | each baseline Glycaemic Status separately. Appendix 8 has the definitions of |
| | | Glycaemic Status at baseline and follow-up. |
| Number of agents for diabetes | 52, 104 | Change from baseline in the total number of medications taken for diabetes defined |
| | | as medications in any of the following classes: metformin, sulphonylurea, |
| | | thiazolidinedione, SGLT-2, GLP-1, and insulin. |
| Proportion of those with diabetes at baseline | 52, 104 | From HbA1c measurement, a binary indicator will be derived, being 1 if participant |
| with HbA1C<7.0% | | achieves the target and 0 if they do not. |
| Proportion of those with diabetes at baseline | 52, 104 | From HbA1c measurement, a binary indicator will be derived, being 1 if participant |
| with HbA1C<6.5% | | achieves the target and 0 if they do not. |
| Change in Albumin-Creatinine Ratio (ACR; | 52, 104 | Follow-up ACR – baseline ACR, only for participants defined as having diabetes, |
| mg/mmol) from baseline for participants | | prediabetes, or hypertension |
| with diabetes, prediabetes, or hypertension | | |
| Obesity-related co-morbidities and their treatments (Hypertension) | ments (Hypertension) | |



| Systolic blood pressure (mmHg) <sup>b</sup> | 52, 104 | Follow-up systolic blood pressure – baseline systolic blood pressure |
|---|---|---|
| ь | 52, 104 | Follow-up diastolic blood pressure – baseline diastolic blood pressure |
| | 52, 104 | Binary indicator of 1 if participant is on antihypertensive medications or systolic |
| | | blood pressure>140mmHg <sup>c</sup> , 0 otherwise with baseline values also presented |
| Number of agents for hypertension | 52, 104 | Change from baseline in total number of medications taken for hypertension |
| | | defined as medications in any of the following classes: ACE-inhibitors, calcium |
| | | channel blockers, thiazide diuretics, alpha-blockers, and beta-blockers. |
| Obesity-related co-morbidities and their treatments (Dyslipidaemia | ents (Dyslipidaemia) | |
| LDL cholesterol (mmol/L) | 52, 104 | Follow-up LDL cholesterol — baseline LDL cholesterol |
| HDL cholesterol (mmol/L) | 52, 104 | Follow-up HDL cholesterol – baseline HDL cholesterol |
| Total cholesterol (mmol/L) | 52, 104 | Follow-up total cholesterol – baseline total cholesterol |
| Triglycerides (mmol/L) | 52, 104 | Follow-up triglycerides – baseline triglycerides |
| Number of agents for dyslipidaemia | 52, 104 | Change from baseline in total number of medications taken for dyslipidaemia defined as medications in any of the following classes: statins, fibrates, and |
| | | ezetimibe. |
| Number of participants referred for other obesity intervention | ity intervention | |
| Referred to Tier 4 for bariatric surgery | 104 | Binary indicator of 1 if participant was referred to Tier 4 for bariatric surgery over 104 week period, 0 otherwise |
| Treatment satisfaction | | |
| Treatment Satisfaction Questionnaire for | 52, 104 | Change from baseline in TSQM scale score. Scored as per version II (detailed in |
| Medication (TSQM) | | Appendix B on vhe 066.fm (iqvia.com). |
| Safety/adverse events | | |
| Gastrointestinal symptoms | 52, 104 | Binary indicator of 1 if participant experienced any nausea or vomiting in study up until the time point of interest (captured in the expected AEs), 0 otherwise |
| Overall hypoglycaemia rate – ADA definition | 52, 104 | Hypoglycaemia events will be defined as per Appendix 5 for people without |



| | | diabetes and as per the ADA definition in Appendix 5 for people with diabetes. |
|---|---|---|
| | | Hypoglycaemia rate will be calculated per participant as total number of |
| | | hypoglycaemia events divided by the total follow-up time. |
| Overall hypoglycaemia rate – Novo Nordisk | 52, 104 | Hypoglycaemia events will be defined as per Appendix 5 for people without |
| definition | | diabetes and as per the Novo Nordisk definition in Appendix 5 for people with |
| | | diabetes. Hypoglycaemia rate will be calculated per participant as total number of |
| | | hypoglycaemia events divided by the total follow-up time. |
| AES | Continual | Defined as in protocol with MEDRA coding used to classify AEs into System Organ |
| | | Classes |
| SAEs | 52, 104 | Defined as in protocol with MEDRA coding used to classify SAEs into System Organ |
| | | Classes |
| Rates of severe hypoglycaemia | 52, 104 | Calculated per participant as total number of severe hypoglycaemia events divided |
| | | by the total follow-up time, where severe hypoglycaemia is defined as |
| | | hypoglycaemic episodes requiring the assistance of another person to actively |
| | | administer carbohydrate, glucagon, or other resuscitative actions (i.e., 'severe |
| | | hypoglycaemic episodes') |
| Change in heart rate from baseline (beats per | 52, 104 | Follow-up heart rate baseline heart rate |
| minute) | | |
| Compliance of patient with the treatment | | |
| Compliant with Tier 3 service (completers) | 52, 104 | Binary indicator of 1 if participant is compliant, 0 otherwise (defined in study |
| Stopped treatment with LIRA 3mg because of | 52, 104 | Binary indicator of 1 if participant stopped treatment with LIRA 3mg because of |
| adverse effects | | |
| | | were currently eligible for LIRA 3mg treatment. * This includes main reason of |
| | | 'adverse event' or 'unable to tolerate drug'. |
| The adherence of participants with the LIRA | 52, 104 | Participants will be defined as treatment compliant if they self-administer at least |
| | | 70% of planned doses. Binary indicator of 1 if participant is compliant, 0 otherwise. |



| baseline calculated. | | (IPAQ- Long Form; MET-minutes/week) |
|---|---|---|
| Total MET-minutes/week calculated in line with Appendix 6 and then change from | 52, 104 | International physical activity questionnaire |
| | | Physical activity assessment |
| Binary indicator of 1 if participant started on anti-obesity drugs other than LIRA 3mg, 0 otherwise. Defined as a concomitant medication listing of Orlistat. | 52, 104 | Started on anti-obesity drugs |
| Binary indicator of 1 if participant completed 52 weeks of the Tier 3 service programme despite stopping LIRA 3mg at 32 weeks, 0 otherwise. Only defined for participants in intervention arm who stopped LIRA 3mg treatment at 32 weeks. | 52 | Completed 52 weeks of Tier 3 service programme despite stopping LIRA 3mg at 32 weeks |
| Binary indicator of 1 if participant completed 52 weeks of the Tier 3 service programme despite stopping LIRA 3mg at 16 weeks, 0 otherwise. Only defined for participants in intervention arm who stopped LIRA 3mg treatment at 16 weeks. | 52 | Completed 52 weeks of the Tier 3 service programme despite stopping LIRA 3mg at 16 weeks |
| Binary indicator of 1 if participant stopped treatment with LIRA 3mg at time-point (i.e., due to stopping rules or side effects), 0 otherwise. Only defined for participants in intervention arm who were on LIRA 3mg treatment at the previous time-point. | 16, 32, 52 | Stopped LIRA 3mg |
| Given the change in visits as a result of COVID-19 to allow face-to-face, this will be defined using the questionnaire answers as detailed in Appendix 7. Only defined for participants in intervention arm who were currently eligible for LIRA 3mg treatment. | | 3mg (monitored through specific questionnaire and return of used pens) |

<sup>&</sup>lt;sup>a</sup> Glucose lowering medications are defined as metformin, a sulphonylurea, a thiazolidinedione, or a SGLT-2.

database. N.B. CPAP compliance (hours/days) was listed as a secondary outcome in the protocol but will not be reported as it hasn't been captured in the

<sup>&</sup>lt;sup>b</sup> These are also considered safety outcomes.

<sup>&</sup>lt;sup>c</sup> On the CRF, hypertension is a yes/no tick box with the following wording: "Hypertension treated (antihypertensives with or without diagnosis) or blockers, thiazide diuretics, alpha-blockers (e.g., doxazosin) and beta-blockers. for the derivation of any variables then the following medication should be considered as anti-hypertensive: ACE-inhibitors, calcium channel untreated (systolic blood pressure >140 mmHG at two consecutive visits to Tier 3 clinic)." If a definition of anti-hypertensive medications is required



# 2.3 Subgroups and/or interactions

No subgroup or interaction analyses are planned.

#### 2.4 Compliance

For assessing the impact of compliance on the effectiveness of the intervention, , compliance is defined as:

Participants in the standard care group are defined as treatment compliant if they complete at least 70% of the planned contacts in the Tier 3 service. Participants in the intervention group are defined as treatment compliant if they complete at least 70% of the planned contacts in the Tier 3 service, and take at least 70% of their planned doses of LIRA 3mg as stipulated by the prescribing pathway.

Compliance variables are listed in Section 2.2.

A binary variable of compliant with tier 3 service captures whether a participant has been compliant with the planned contacts in Tier 3 service (see section 3.3.3).

#### 2.5 Other

There are no other variables to be presented in the statistical report which are not outcomes, baseline or demographic variables, or for measuring compliance or safety.

Trial:

**STRIVE** SAP Version: 1.1 DRAFT

Version Date: 01/08/2022



# **Analysis Sets/Populations**

# 3.1 Disposition of participants

#### **Screened patients**

Screened patients are defined as any patient who met the inclusion criteria and signed the informed consent form.

#### **Treated patients**

Treated patients consist of all patients, who have been allocated to one of the two treatment groups, and have at least partially completed the Baseline Visit.

Data from all randomised participants will be used in the study final report and analysis, with data analysed in the group to which the participant was randomised.

#### 3.2 Protocol deviations

The following deviations were captured in the protocol deviation Case Report Form:

| Participant ineligible for entry into trial | |
|------------------------------------------------|-----------------|
| Participant deviated from randomised treatment | ent group |
| Participant's visit/assessment not performed | as per protocol |
| Non-permitted treatment | |
| Trial Specific Issues | - |
| Other deviation | |

No protocol deviations will result in systematic exclusion from all statistical analyses. Reasons for exclusion/inclusion in each population are described in 3.3. below.

#### 3.3 Populations

All treated patients will be included in the Intention-To-Treat (ITT) population as a minimum. Patients who were screened, but not treated, will not be included in any of the analysis populations.

# 3.3.1 Complete Cases Population

The complete cases population is defined as all randomised participants who have data available for the outcome being analysed, according to the study group to which they were randomised at baseline. Participants who had bariatric surgery during the study period will be only be included at time-points prior to their bariatric surgery. They will be excluded from time-points after their bariatric surgery.



#### 3.3.2 Intention-To-Treat Population

The ITT population are all randomised participants and they will be analysed according to the treatment group to which they were randomised at baseline.

Missing outcome data will be imputed. Participants who had bariatric surgery during the study period will be included in this population.

Missing primary outcome data will need to be imputed for the ITT analyses; this will be done by assuming that these participants did not achieve ≥15% weight loss at 52 weeks, which is a conservative approach.

#### 3.3.3 Per Protocol Population

The per protocol population is defined as all participants who were compliant with their randomised treatment group, analysed according to the treatment group to which they have randomised at baseline. Participants in the standard care group are defined as treatment compliant if they complete at least 70% of the planned contacts in the Tier 3 service. Participants in the intervention group are defined as treatment compliant if they complete at least 70% of the planned contacts in the Tier 3 service, and take at least 70% of their planned doses of LIRA 3mg as stipulated by the prescribing pathway.

Participants that had Liraglutide 3mg outside of the treatment pathway (i.e. in the control group or in the intervention group after a stopping rule means they should have stopped taking Liraglutide 3mg) will be excluded from the per protocol population. The protocol deviations and in particular deviations from randomised treatment group in the protocol deviations will capture where this has occurred for any individual.

Participants who had bariatric surgery during the study period will be only be included at time-points prior to their bariatric surgery. They will be excluded from time-points after their bariatric surgery.

The binary variable of compliant with tier 3 service at 52 weeks will be used to exclude individuals that did not have 70% of planned visits for outcomes assessed at 52 weeks, likewise for outcomes assessed at 104 weeks the variable at 104 weeks will be used.

Individuals in the intervention arm that did not receive 70% of the doses as determined by the protocol (i.e. in the first 16 weeks or there after whilst continuing to meet the continue rules of the protocolised treatment schedule) will be excluded from the per protocol populations. The number of days taking LIRA and whether this corresponds to 70% of doses is defined in Appendix 7 in section 14. For outcomes at



the 52 week time point the definition in 14.1 should be used; while for outcomes at the 104 week time point the definition in 14.2 should be used.

#### 3.3.4 Responder Population

The Responder population is defined as all participants in the intervention group who achieved ≥15% weight loss at 52 weeks, and all participants in the standard care group. Participants will be analysed according to the treatment group to which they were randomised at baseline.

Participants who had bariatric surgery during the study period will be only be included at time-points prior to their bariatric surgery. They will be excluded from time-points after their bariatric surgery.

#### 3.3.5 Safety Population

All individuals randomised into the trial will be in the safety population. Individuals randomised to the intervention will be analysed in the intervention arm unless they have not receive a dose of LIRA on the prescribed treatment pathway i.e. the protocol deviations and in particular a deviation from randomised treatment group indicates this is the case. Individuals randomised to the control arm will be analysed in the control arm unless they have received a dose of LIRA as part of the prescribed treatment pathway i.e. the protocol deviations and in particular a deviation from randomised treatment group indicates this is the case.



# 4 General Issues for Statistical Analysis

#### 4.1 Analysis Groups

In all analyses, participants will be analysed in the group to which they were randomised at baseline; importantly, the participants in the intervention group who stop LIRA 3mg, because they meet a pre-specified stopping rule, will still be analysed in the intervention group.

#### 4.2 Missing Data

Attempts will be made to assess the primary outcome on all participants including those who have withdrawn from treatment. The number of missing observations for each outcome will be reported. If missing outcome data are present then the initial analysis will be based on the complete cases. A sensitivity analysis will then be carried out repeating the analyses with the ITT population to assess the possible impact of the missing data on the results produced. Missing primary outcome data will need to be imputed for the ITT analyses; this will be done by assuming that these participants did not achieve ≥15% weight loss at 52 weeks, which is a conservative approach. We will also attempt to address bias by comparing the characteristics of those with missing outcome data to those who have completed follow-up. This strategy for dealing with missing outcome data has been recommended by White et al. (White 2011)

There should be no missing covariate data because site and baseline BMI are used as part of the randomisation process. The other covariate is treatment group which was assigned as part of the randomisation process and will be known for all participants.

Where participants were lost to follow up or missed a study visit, the study team attempted to access primary outcome data from existing hospital, GP or health records, where appropriate consent was in place.

# 4.3 Derived/Computed Variables

Analyses will be adjusted for the stratification variables which are study site and body mass index (BMI).

Study site is a non-ordinal, categorical, dummy variable with a unique code for each site.

BMI is a continuous variable calculated as weight in kg divided by height in metres squared. For stratification purposes, baseline BMI was dichotomised based on cut-off values of  $\geq$ 45kg/m<sup>2</sup> and <45kg/m<sup>2</sup>. This dichotomised grouping will be included in statistical models.



# 4.4 Multiple Testing

No corrections will be made for multiple testing. However, due to the large amount of secondary outcomes, statistical models will only be fitted for the most important secondary outcomes to limit the impact of multiple testing. Descriptive summaries will be produced for the other secondary outcomes without multiple testing, as described below.

# 4.5 Analysis Software

Latest version of Stata, SAS, or other appropriate statistical software.

# 4.6 Statistical Significance

All statistical tests, p-values, and confidence intervals will be two-sided. Statistical significance will be assessed at the 5% level for main effects. No interaction analyses are planned, however if post-hoc interaction effects are tested then these will be assessed at the 10% level.

#### 4.7 Outliers

Given that the study participants are taking part in this study because of issues around weight control, outliers will not be removed from the dataset as these could feasibly be genuine extremes.



# 5 Statistical Methodology

#### 5.1 Disposition

A CONSORT diagram showing the flow of participants through the study will be produced, including the number of screened and treated participants. This diagram will also show the number of participants receiving the allocated treatment at each stage of the study, along with the reasons for stopping treatment. In particular, the number who stop LIRA 3mg due to each stopping rule will be clearly stated.

The number (percentage) of participants in each analysis population will be tabulated overall and by treatment group. The type and number (percentage) of protocol deviations will also be tabulated overall and by treatment group in the ITT population.

# 5.2 Interim analysis

No interim analysis is planned.

# 5.3 Demographic and Baseline Characteristics

Baseline characteristics of the participants will be summarised by randomisation group and overall using mean (standard deviation) and median (interquartile range) for continuous variables and count (percentage) for categorical variables. There will be no tests of statistical significance nor confidence intervals for differences between randomised groups on any baseline variable.

Additionally, the baseline characteristics of those with missing primary outcome data will be summarised separately from those with complete primary outcome data using mean (standard deviation) and median (interquartile range) for continuous variables and count (percentage) for categorical variables. These characteristics will be compared using a t-test for normally distributed variables, a Mann-Whitney test for non-normally distributed variables, and a chi-squared test for categorical variables.

# 5.4 Primary Outcome Analysis

The complete cases, ITT, and per protocol analyses will compare the two groups to demonstrate the effectiveness of the targeted prescribing pathway compared with standard care.



#### 5.4.1 Primary Analysis of Primary Outcome

The primary analysis will compare the proportion of participants achieving  $\geq 15\%$  weight loss at 52 weeks (primary outcome) after randomisation between the two randomisation groups. The primary outcome will be summarised using count and percentage. A logistic regression model will be used with a binary indicator showing whether or not  $\geq 15\%$  weight loss was achieved at 52 weeks as the outcome, randomisation group (intervention or control) as the main covariate, and the stratification factors of site (non-ordinal categorical variable) and baseline BMI ( $\geq 45 \text{kg/m}^2$ ;  $< 45 \text{kg/m}^2$ ) as additional covariates. The adjusted odds ratio will be presented, 95% confidence interval and p-value comparing the two groups.

The primary analysis will use the complete cases population, therefore missing data will not be imputed.

#### 5.4.2 Secondary Analyses of Primary Outcome

The primary analysis of the primary outcome will be repeated using the ITT and per protocol populations as secondary analyses. Missing primary outcome data will need to be imputed for the ITT analyses; this will be done by assuming that these participants did not achieve ≥15% weight loss at 52 weeks, which is a conservative approach.

#### 5.4.3 Sensitivity Analyses

No sensitivity analyses are planned.

#### 5.4.4 Exploratory Analyses

The per-protocol analysis of the primary outcome will be repeated in the per-protocol population but also excluding individuals had any of the following concomitant medications before their 52 week weight measure was recorded:

- Orlistat
- GLP-1 at glucose lowering dose
- Bupropion/Naltrexone
- SGLT-2 inhibitor which was started after randomisation

#### 5.5 Secondary Outcome Analyses

#### 5.5.1 Primary Analysis of Secondary Outcomes

Secondary anthropometric outcomes will be analysed in a similar way to the primary analysis. These outcomes will be summarised overall and by treatment group.



Categorial outcomes will be summarised using count and percentage. Continuous outcomes will be summarised using mean, standard deviation, median, range, and interquartile range. Binary anthropometric outcomes will be compared between the two treatment arms using logistic regression models with the anthropometric outcome as the outcome and randomisation group and the stratification factors (site, baseline BMI) as covariates. The adjusted odds ratio will be presented along with 95% confidence interval and p-value comparing the two treatment arms. Continuous anthropometric outcomes will be compared using linear regression models with the anthropometric outcome as the outcome and randomisation group and the stratification factors (site, BMI) as covariates. The adjusted mean difference will be estimated along with 95% confidence interval and p-value comparing the two treatment arms. If continuous outcomes are non-normally distributed then they will be transformed or a more suitable regression model will be selected.

No formal statistical testing will take place for the other secondary outcomes due to the large amount of secondary outcomes and to reduce multiple testing. Instead, descriptive analyses will be performed to explore potential patterns in improvements. This will apply to the outcomes relating to obesity-related co-morbidities, referrals to Tier 4 services, treatment satisfaction, treatment compliance, and physical activity. Categorial outcomes will be summarised using count and percentage. Continuous outcomes will be summarised using mean, standard deviation, median, range, and interquartile range. Where it makes sense to do so, for continuous variables the baseline, follow-up, and change values will all be summarised; some outcomes can only be defined at follow-up and so this will not apply to those outcomes.

In all analyses, participants will be analysed in the group to which they were randomised at baseline. Only the complete cases population will be used for the secondary outcomes to reduce the number of models being fitted. Participants who have undergone bariatric surgery during the period of the study will be excluded from these analyses if their bariatric surgery took place before the analysed time-point.

#### 5.5.2 Secondary Analyses of Secondary Outcomes

As additional secondary analyses, we will perform a responder analysis which will repeat the analyses of the secondary anthropometric outcomes with the intervention group restricted to those participants who responded to the targeted prescribing pathway (i.e. had achieved ≥15% weight loss at 52 weeks after randomisation). The purpose of these analyses is to compare the outcomes of "early and good" responders to the targeted prescribing pathway with those who received standard care only.



Therefore, all participants randomised to the standard care group will also be included in these responder analyses.

#### 5.5.3 Sensitivity Analyses

No sensitivity analyses are planned.

#### 5.6 Subgroup Analyses

No subgroup analyses are planned.

# 5.7 Figures to be produced

| Figure | Description |
|---|---|
| CONSORT diagram | See Section 5.1 |
| Treatment flow | Based on figure in Section 1.2.1 with numbers added to show number of participants at each stage |

# 5.8 Changes to the Planned Analysis

In the protocol, it stated that most secondary outcomes would be subject to formal statistical testing, with some secondary outcomes (safety, treatment compliance, treatment satisfaction) tabulated only, without statistical testing. However, due to the large number of secondary outcomes, it was decided that more secondary outcomes should be tabulated only to reduce the impact of multiple testing. The following outcomes were the ones for which the approach changed: obesity-related comorbidities, referrals to Tier 4 services, and physical activity.

In the protocol, the majority of the secondary outcomes were listed as absolute values, however the change from baseline will instead be analysed for continuous variables.

In the protocol, it states that ACR will be analysed as a secondary outcome for participants with diabetes. However, ACR was also measured for participants with prediabetes or hypertension and so these have been added to the ACR secondary outcome definition.

In the protocol, it was stated that participants who had bariatric surgery would be excluded from the complete cases, per protocol, and responder populations. However, it is more likely that these individuals will be poor responders and so excluding them could potentially bias the analyses. Therefore, participants who had bariatric surgery during the study period will be only be included at time-points prior to their bariatric surgery. They will be excluded from time-points after their bariatric surgery.



In the protocol, it stated that adjusted proportions or means would be presented by treatment group in the primary and secondary analyses. However, the unadjusted raw values are presented instead.


### 6 Safety and Adverse events (AEs)

The safety outcomes (including AEs and SAEs) will be summarised overall, by randomisation group, and by whether or not the participant was currently receiving LIRA 3mg treatment using count and percentage. The following information will also be presented:

- Incidence rate (per person-year) of each System Organ Class of AEs by treatment and overall
- Proportion of participants with at least one AE, by System Organ Class type, treatment arm, and overall
- Incidence rate (per person-year) of each expected AE type by treatment and overall
- Proportion of participants with at least one expected AE, by AE type, treatment arm, and overall
- Bar chart of number of AEs per individual, split by treatment
- Proportion of individuals with at least one AE of given severity by treatment and overall
- Proportion of individuals with at least one AE of given 'likelihood related' by treatment and overall.

For System Organ Classes with >0.1 AEs per person-year, the AEs broken down by higher level term.

Additionally, separate listings of all AEs and SAEs will be produced, including 'likelihood related', expectedness, duration, severity, action taken, outcome, and treatment, with sorting by randomisation group, participant ID, then date.

Finally, hypogylcaemia events will be tabulated by Glycaemic status for ADA and Novo Nordisk definition separately.

The safety analyses will use the safety population.



### 7 References

White IR, Horton NJ, Carpenter J, Pocock SJ. Strategy for intention to treat analysis in randomised trials with missing outcome data. BMJ. **2011**;342:d40.



### 8 Appendix 1: Scoring for King's College Obesity Staging System

| | Stage 0 | Stage 1 | Stage 2 | Stage 3 |
|---|---|---|---|---|
| | Normal Health | At risk of disease | Established disease | Advanced disease |
| Airways | Normal | Snoring | CPAP therapy | Cor pulmonale |
| ВМІ | <35kg/m <sup>2</sup> | 35-40 kg/m <sup>2</sup> | 40-60 kg/m <sup>2</sup> | >60 kg/m <sup>2</sup> |
| Cardiovascular | <10% risk | 10-20% risk | Heart disease | Heart failure |
| Diabetes | Normal | Impaired fasting glucose | Type 2 diabetes | Uncontrolled type 2<br>diabetes |
| Economic | Normal | Increased expense<br>for clothes and<br>travel | Workplace<br>discrimination | Unemployment due to obesity |
| Functional | Can walk three flights of stairs | Can walk one or two flights of stairs | Requires mobility aid | Housebound |
| Gonadal | Normal | PCOS/erectile<br>dysfunction | Subfertility | Sexual dysfunction leading to relationship breakdown |
| Health status (perceived) | Normal | Low mood or QoL | Depression or poor<br>QoL | Severe depression |
| Image (body) | Normal | Dislikes body | Body image<br>dysphoria | Eating disorder |

Abbreviations: CPAP, Continuous Positive Airway Pressure; PCOS, Polycystic Ovarian Syndrome; QoL, Quality of Life.



### 9 Appendix 2: Scoring for PHQ-9 Questionnaire

### PHQ-9\* Questionnaire for Depression Scoring and Interpretation Guide

### For physician use only

Count the number (#) of boxes checked in a column. Multiply that number by the value indicated below, then add the subtotal to produce a total score. The possible range is 0-27. Use the table below to interpret the PHQ-9 score.

| Not at all | (#) x 0 = |
|-------------------------|-----------|
| Several days | (#) x 1 = |
| More than half the days | (#) x 2 = |
| Nearly every day | (#) x 3 = |
| Total coores | |

| | | Interpretin | g PHQ-9 Scores |
|---|---|---|---|
| Diagnosis | Total Score | For Score | Action |
| Minimal depression | 0-4 | ≤4 | The score suggests the patient may not need depression treatment |
| Mild depression<br>Moderate depression | 5-9<br>10-14 | 5 - 14 | Physician uses clinical judgment about treatment, based on patient's duration of symptoms and functional impairment |
| Moderately severe depression<br>Severe depression | n 15-19<br>20-27 | > 14 | Warrants treatment for depression, using antidepressant, psychotherapy and/or a combination of treatment. |



### 10 Appendix 3: Scoring for Epworth Sleepiness Scale

### **How Sleepy Are You?**

How likely are you to doze off or fall asleep in the following situations? You should rate your chances of dozing off, not just feeling tired. Even if you have not done some of these things recently try to determine how they would have affected you.

For each situation, decide whether or not you would have:

- No chance of dozing =0
- · Slight chance of dozing =1
- Moderate chance of dozing =2
- High chance of dozing =3

Write down the number corresponding to your choice in the right-hand column. Total your score below.

### **Situation Chance of Dozing**

Sitting and reading ·

Watching TV ·

Sitting inactive in a public place (e.g., a theater or a meeting) ·

As a passenger in a car for an hour without a break ·

Lying down to rest in the afternoon when circumstances permit ·

Sitting and talking to someone ·

Sitting quietly after a lunch without alcohol ·

In a car, while stopped for a few minutes in traffic ·

| ı | ota | 13 | CO | re | = |
|---|-----|----|----|----|---|

### **Analyze Your Score**

### Interpretation:

≥10: Requires referral for sleep apnoea studies as indicates above average daily sleepiness.



### 11 Appendix 4: Scoring for Stop Bang Questionnaire

| 1. | Do you <b>Snore</b> loudly? Louder than talking or loud enough to be heard through a closed door | Yes | No |
|---|---|---|---|
| 2. | Has anybody Observed you stop breathing during your sleep? | Yes | No |
| 3. | Do you often feel <b>Tired</b> , fatigued, or sleepy during the daytime? | Yes | No |
| 4. | High Blood Pressure? – do you have it or are you on treatment? | Yes | No |
| 5. | Gender: Are you male or female? | М | F |
| 6. | Is your <b>Age</b> above 50? | Yes | No |

| cm / | Ni ala da a da a da a da a da a da a da a | 1 | |
|--------|-------------------------------------------|-------------|----|
| ( ) | Neck circumference | Yes | No |
| inches | >40cm? | | |
| kg | - | - | = |
| m | - | - | - |
| kg/m2 | BMI > 35 kg/m2 | Yes | No |
| | kg<br>m | kg -<br>m - | kg |

If the **STOP-BANG** score is **5** or more, consideration should be given to referral to the Sleep Service for investigation and treatment of possible Obstructive Sleep Apnoea (OSA).

- A score of 3 or more is sensitive for moderate-severe OSA but is not very specific, there is a high false positive rate.
- A score of 5-8 is far more specific and indicates a high probability of moderatesevere OSA.



### 12 Appendix 5: Definitions of hypoglycaemia

A hypoglycaemic episode will be defined as treatment emergent if the onset of the episode is on or after the first day of randomised treatment and no later than 14 days after the last day of randomised treatment. Hypoglycaemic events will be defined as nocturnal if the time onset is between 00:01 and 05:59 (both included).

A hypoglycaemic episode form and an Adverse Event (AE) form must be filled in for all hypoglycaemic episodes. Hypoglycaemic episodes requiring the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions (i.e., 'severe hypoglycaemic episodes') will be qualified as an event of special interest.

A different definition of hypoglycaemia will apply for patients with type 2 diabetes and a different definition will apply for patients without diabetes.

### Classification of hypoglycaemia for participants with type 2 diabetes

All participants with diabetes will be supplied with a glucose meter and a diabetes diary for recording of hypoglycaemia, symptomatic episodes and routine blood glucose monitoring. Plasma glucose should always be measured from all participants with diabetes when there is the suspicion of a hypoglycaemic episode.

All plasma glucose values ≤3.1 mmol/L (56mg/dL), as well as values >3.1 mmol/L (56mg/dL) when hypoglycaemic symptoms have occurred should be recorded by the participants in the diaries. Hypoglycaemic episodes will be recorded by the participant in his/her diary throughout the trial and must be transcribed into the CRF by the Investigator at each site visit throughout the trial.

Hypoglycaemic episodes will be summarised based on the American Diabetes Association (ADA) classification and Novo Nordisk's definition.

### **Novo Nordisk definition**

In normal physiology, hypoglycaemia symptoms occur at a blood glucose level of approximately < 2.8 mmol/L (50 mg/dL)/plasma glucose level < 3.1 mmol/L (56 mg/dL). Therefore, Novo Nordisk has used this cut-off value to define minor hypoglycaemia.

Minor hypoglycaemic episode is defined as:

 An episode with symptoms consistent with hypoglycaemia with confirmation by plasma glucose < 3.1 mmol/L (56 mg/dL), or full blood glucose < 2.8 mmol/L (50 mg/dL) and which is handled by the subject himself/herself



• Or any asymptomatic plasma glucose value < 3.1 mmol/L (56 mg/dL) or full blood glucose value < 2.8 mmol/L (50 mg/dL). Minor hypoglycaemic episodes will be summarised according to this definition, and can be subject to additional analysis.

### **ADA hypoglycaemia classification**

According to ADA the definition of a hypoglycaemic episode is categorised as:

<u>Severe hypoglycaemia:</u> An episode requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions.

<u>Documented symptomatic hypoglycaemia:</u> An episode during which typical symptoms of hypoglycaemia are accompanied by a measured plasma glucose concentration ≤3.9 mmol/L.

<u>Asymptomatic hypoglycaemia:</u> An episode not accompanied by typical symptoms of hypoglycaemia, but with a measured plasma glucose concentrations ≤3.9 mmol/L.

<u>Probable symptomatic hypoglycaemia:</u> An episode during which symptoms of hypoglycaemia are not accompanied by a plasma glucose determination (but that was presumably caused by a plasma glucose concentration ≤3.9mmol/L).

Relative hypoglycaemia: An episode during which the participant reports any of the typical symptoms of hypoglycaemia and interprets those as indicative of hypoglycaemia, but with a measured plasma glucose concentration >3.9 mmol/L.

### <u>Classification of hypoglycaemia for participants without diabetes</u>

Participants without diabetes will not be routinely provided with blood glucose meters or diaries; hence blood glucose will not be measured in case of symptoms of hypoglycaemia unless it coincides with a clinic visit.

The hypoglycaemia events for participants without diabetes will be reported spontaneously i.e., symptoms of hypoglycaemia (not biochemically confirmed) occurring outside of visits to the clinic; severe hypoglycaemia will be defined as an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. In the event of severe or symptomatic hypoglycaemia patients will be given a glucose monitor and asked to record their blood glucose whenever they feel symptomatic.



### 13 Appendix 6: IPAQ scoring system

Further details including data processing rules can be found here: https://sites.google.com/site/theipaq/scoring-protocol

### **Continuous Score**

Data collected with the IPAQ long form can be reported as a continuous measure and reported as median MET-minutes. Median values and interquartile ranges can be computed for walking (W), moderate-intensity activities (M), and vigorous-intensity activities (V) within each domain using the formulas below. Total scores may also be calculated for walking (W), moderate-intensity activities (M), and vigorous-intensity activities (V); for each domain (work, transport, domestic and garden, and leisure) and for an overall grand total.

### **MET Values and Formula for Computation of MET-minutes**

### **Work Domain**

Walking MET-minutes/week at work = 3.3 \* walking minutes \* walking days at work Moderate MET-minutes/week at work = 4.0 \* moderate-intensity activity minutes \* moderate-intensity days at work

Vigorous MET-minutes/week at work= 8.0 \* vigorous-intensity activity minutes \* vigorous-intensity days at work

Total Work MET-minutes/week = sum of Walking + Moderate + Vigorous MET-minutes/week scores at work.

### **Active Transportation Domain**

Walking MET-minutes/week for transport = 3.3 \* walking minutes \* walking days for transportation

Cycle MET-minutes/week for transport= 6.0 \* cycling minutes \* cycle days for transportation

Total Transport MET-minutes/week = sum of Walking + Cycling MET-minutes/week scores for transportation.

### **Domestic and Garden [Yard Work] Domain**

Vigorous MET-minutes/week yard chores = 5.5 \* vigorous-intensity activity minutes \* vigorous-intensity days doing yard work (Note: the MET value of 5.5 indicates that vigorous garden/yard work should be considered a moderate-intensity activity for scoring and computing total moderate intensity activities.)

Moderate MET-minutes/week yard chores= 4.0 \* moderate-intensity activity minutes \* moderateintensity days doing yard work



Moderate MET-minutes/week inside chores = 3.0\* moderate-intensity activity minutes \* moderateintensity days doing inside chores.

Total Domestic and Garden MET-minutes/week =sum of Vigorous yard + Moderate yard + Moderate inside chores MET-minutes/week scores.

### **Leisure-Time Domain**

Walking MET-minutes/week leisure = 3.3 \* walking minutes \* walking days in leisure Moderate MET-minutes/week leisure = 4.0 \* moderate-intensity activity minutes \* moderate-intensity days in leisure

Vigorous MET-minutes/week leisure = 8.0 \* vigorous-intensity activity minutes \* vigorous-intensity days in leisure

Total Leisure-Time MET-minutes/week = sum of Walking + Moderate + Vigorous MET-minutes/week scores in leisure.

### Total Scores for all Walking, Moderate and Vigorous Physical Activities

Total Walking MET-minutes/week = Walking MET-minutes/week (at Work + for Transport + in Leisure)

Total Moderate MET-minutes/week total = Moderate MET-minutes/week (at Work + Yard chores + inside chores + in Leisure time) + Cycling Met-minutes/week for Transport + Vigorous Yard chores MET-minutes/week

Total Vigorous MET-minutes/week = Vigorous MET-minutes/week (at Work + in Leisure)

Note: Cycling MET value and Vigorous garden/yard work MET value fall within the coding range of moderate-intensity activities.

### **Total Physical Activity Scores**

An overall total physical activity MET-minutes/week score can be computed as: Total physical activity MET-minutes/week = sum of Total (Walking + Moderate + Vigorous) METminutes/week scores.

This is equivalent to computing: Total physical activity MET-minutes/week = sum of Total Work + Total Transport + Total Domestic and Garden + Total Leisure-Time MET-minutes/week scores.

As there are no established thresholds for presenting MET-minutes, the IPAQ Research Committee proposes that these data are reported as comparisons of median values and interquartile ranges for different populations.



### 14 Appendix 7 Definitions for adherence of participants with the LIRA 3mg

Individuals that didn't receive 70% of the doses as determined by the protocol (i.e. in the first 16 weeks or there after whilst continuing to meet the continue rules of the protocolised treatment schedule) will be classed as not adhering with the LIRA 3mg pathway.

### Defining days taking LIRA

The number of days taking LIRA will be calculated as the time from first dose dispensed (normally at baseline visit) to the last known date of individuals taking the LIRA. Where individuals are recorded as not completing the trial due to stopping the LIRA, the date of last dose of LIRA in the completion form will be used; if this is not recorded then the date of first visit at which individuals say they are not happy to continue taking LIRA will be used; and where neither of these are recorded the date of the last visit that individuals said they are happy to continue LIRA will be used.

### 14.1 52 weeks

Individuals will then be assessed for whether they have received 70% as per table below.

| Delow. | | |
|---|---|---|
| Stopping rule on | Did not receive 70% of | Did receive 70% of |
| protocolised treatment | planned doses | planned doses |
| schedule | | |
| Did not meet rule to | If days taking LIRA is | If days taking LIRA is |
| continue on Lira at 16 | < 70% of days between | ≥70% of days between |
| weeks (either <5% weight | baseline and Week 16. | baseline and Week 16. |
| loss or not measured) | Or, if Week 16 date | Or, if Week 16 date |
| | missing, if days taking | missing, if days taking |
| | LIRA is $\leq$ 78. | LIRA is >78 |
| Did meet rule to continue | If days taking LIRA is | If days taking LIRA is |
| Lira (≥5% weight loss) at | <70% of days between | ≥70% of days between |
| 16 weeks but did not meet | baseline and Week 32. | baseline and Week 32. |
| rule to continue Lira at 32 | Or, if Week 32 date | Or, if Week 32 date |
| weeks (either <10% weight | missing, if days taking | missing, if days taking |
| loss or not measured) | LIRA is ≤156. | LIRA is >156. |
| Did meet rule to continue | If days taking LIRA is | If days taking LIRA is |
| Lira (≥5% weight loss) at | <70% of days between | ≥70% of days between |
| 16 weeks and did meet rule | baseline and week 52. | baseline and week 52. |
| to continue Lira at 32 | Or, if week 52 date | Or, if week 52 date is |
| weeks (≥10% weight loss) | missing, if days taking | missing, if days taking |
| | LIRA is ≤254. | LIRA is >254. |



### 14.2 104 weeks

Individuals will then be assessed for whether they have received 70% as per table below.

| DEIOW. | | TELEVISION TO THE PROPERTY OF |
|---|---|---|
| Stopping rule on | Did not receive 70% of | Did receive 70% of |
| protocolised treatment | planned doses | planned doses |
| schedule | | |
| Did not meet rule to | If days taking LIRA is | If days taking LIRA is |
| continue on Lira at 16 | <70% of days between | ≥70% of days between |
| weeks (either <5% weight | baseline and Week 16. | baseline and Week 16. |
| loss or not measured) | Or, if Week 16 date | Or, if Week 16 date |
| | missing, if days taking | missing, if days taking |
| | LIRA is $\leq$ 78. | LIRA is >78 |
| Did meet rule to continue | If days taking LIRA is | If days taking LIRA is |
| Lira (≥5% weight loss) at | <70% of days between | ≥70% of days between |
| 16 weeks but did not meet | baseline and Week 32. | baseline and Week 32. |
| rule to continue Lira at 32 | Or, if Week 32 date | Or, if Week 32 date |
| weeks (either <10% weight | missing, if days taking | missing, if days taking |
| loss or not measured) | LIRA is ≤156. | LIRA is >156. |
| Did meet rule to continue | If days taking LIRA is | If days taking LIRA is |
| Lira (≥5% weight loss) at | <70% of days between | ≥70% of days between |
| 16 weeks, did meet rule to | baseline and week 52. | baseline and week 52. |
| continue Lira at 32 weeks | Or, if Week 52 date | Or, if Week 52 date |
| (≥10% weight loss) and | missing, if days taking | missing, if days taking |
| did not meet rule to | LIRA is ≤254. | LIRA is >254. |
| continue Lira at 52 weeks | | |
| (either <15% weight loss | | |
| or not measured) | | |
| Did meet rule to continue | If days taking LIRA is | If days taking LIRA is |
| Lira (≥5% weight loss) at | <70% of days between | ≥70% of days between |
| 16 weeks, did meet rule to | baseline and week 104. | baseline and week 104. |
| continue Lira at 32 weeks ( | Or, if Week 104 date | Or, if Week 104 date |
| ≥10% weight loss) and did | missing, if days taking | missing, if days taking |
| meet rule to continue Lira | LIRA is ≤510. | LIRA is >510. |
| at 52 weeks (≥15% weight | _ | |
| loss) | 320 | |
| · | L.,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | |



### 15 Appendix 8: Baseline and follow-up Glycaemic Status Definitions

### 15.1 Baseline Glycaemic Status

Individuals are classified as having diabetes remission status if all of the following is the satisfied:

 HbA1C <6.5%, not on glucose lowering medication and have a previous medical history of diabetes

Individuals are classified as having diabetes status if one of the following is the satisfied:

- HbA1C ≥6.5%
- Have previous medical history of diabetes and they are on any glucose lowering medication (including Metformin)
- Are on any glucose-lowering medication except of Metformin (with or without past medical history of diabetes).

Individuals are classified as having pre-diabetes status if one of the following is the satisfied:

- HbA1C 6.0-6.4%, without a previous medical history of diabetes and not on any glucose-lowering medication.
- HbA1C 6.0-6.4%, without a previous medical history of diabetes and only on Metformin from glucose-lowering medications.
- HbA1C <6.0%, with a previous medical history of pre-diabetes (but without a previous medical history of diabetes) and only on Metformin from glucoselowering medications.

Individuals are classified as having Normoglycaemia if one of the following is satisfied:

- HbA1C <6.0%, without a previous medical history of diabetes and not on any glucose-lowering medication.
- HbA1C <6.0%, without a previous medical history of diabetes or pre-diabetes and only on Metformin from glucose-lowering medications.



### 15.2 Follow-up Glycaemic Status

Individuals are classified as having diabetes remission status if all the following is satisfied:

 Follow-up HbA1C <6.5%, not on glucose lowering medication for ≥ 3months, have a previous medical history of diabetes and have NOT being on LIRA 3mg within the last 3 months

Individuals are classified as having diabetes status if one of the following is the satisfied:

- Follow-up HbA1C ≥6.5%
- Have previous medical history of diabetes and they are on any glucose lowering medication (including Metformin) within the last 3 months and/or have being on LIRA 3mg within the last 3 months
- Are on any glucose-lowering medication except of Metformin (LIRA 3mg is considered obesity medication, not glucose-lowering)

Individuals are classified as having pre-diabetes status if one of the following is the satisfied:

- Follow-up HbA1C 6.0-6.4%, without previous medical history of diabetes and not on any glucose-lowering medication (but they can be on LIRA 3mg).
- Follow-up HbA1C 6.0-6.4%, without previous medical history of diabetes and only on Metformin from glucose lowering agents (and they can also be on LIRA 3mg).
- Follow-up HbA1C <6.0%, with a previous medical history of pre-diabetes (but without a previous medical history of diabetes) and only on Metformin from glucose-lowering agents (and they can also be on LIRA 3mg).

Individuals are classified as having Normoglycaemia if one of the following is the satisfied:

- Follow-up HbA1C <6.0%, without a previous medical history of diabetes and not on any glucose-lowering medication (but they can be on LIRA 3mg).
- Follow-up HbA1C <6.0%, without a previous medical history of diabetes or prediabetes and only on Metformin from glucose-lowering medications (and they can also be on LIRA 3mg).



### 16 Appendix 9: Templates for Tables

### 16.1 Disposition

| Population | | rol group<br>n = ) | | tion group<br>1 = ) | The Contract of the Contract o | opulation<br>n = ) |
|---|---|---|---|---|---|---|
| | Number | Percentage | Number | Percentage | Number | Percentage |
| Complete cases | | | | | | |
| Intention-to-treat | | | | | | |
| Of whom, those who had bariatric surgery | | | | | | |
| Per protocol | | | | | | |
| Responder | | | | | | |

### 16.2 Protocol deviations

| Type of protocol | | rol group<br>n = ) | | tion group<br>n = ) | | opulation<br>n = ) |
|---|---|---|---|---|---|---|
| deviation | Number | Percentage | Number | Percentage | Number | Percentage |
| [TBC] | | | | | | |
| [TBC] | | | | | | |
| [TBC] | | | | | | |
| [TBC] | | | | | | |



## 16.3 Summary of continuous baseline characteristics

| | | Control group<br>(n = ) | trol grou<br>(n = ) | d | | | Intervention group<br>(n = ) | ention g<br>(n = ) | roup | | | Tota | | Total population<br>(n = ) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Baseline characteristic | N missing | Mean | SD | Median | IQR | N<br>missing | Mean | SD | Median | IQR | N<br>missin | 5 | n Mean | - |
| Age, years | | | | | | | | | | | | | | |
| Weight, kg | | | | | | | | | | | | | | |
| Body mass index, kg/m <sup>2</sup> | | | | | | | | | | | | | | |
| Heart rate, beats/minute | | | | | | | | | | | | - | | |
| Waist circumference, cm | | | | | | | | | | | | | | |
| HbA1c, mmol/mol | | | | | | | | | | | | - | | |
| HbA1c, % | | | | | | | | | | | | | | |
| Albumin-creatinine ratio, | | | | | | | | | | | | | | |
| mg/mmol | | | | | | | | | | | | | | |
| Systolic blood pressure, | | | | | | | | | | | | | | |
| mmHg | | | | | | | | | | | | | | |
| Diastolic blood pressure, | | | | | | | | | | | | | | |
| mmHg | | | | | | | | | | | | | | |
| LDL cholesterol, mmol/L | | | | | | | | | | | | | | |



| | | Control group | ol grou | ē | | | Intervention group | tion g | roup | | | Tota | Total population $(n = 1)$ | ion | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n) | (n = ) | | | | (1 | (n = ) | | | | | (n = ) | | |
| Baseline characteristic N missing | N missing | Mean | SD | SD Median IQR | Я | N N SD Median IQR missin Mean | Mean | SD | Median | iQR | missin<br>g | | SD | Median | ō |
| HDL cholesterol, mmol/L | | | | | | | | | | | | | | | |
| Total cholesterol, mmol/L | | | | | | | | | | | | | | | |
| Triglycerides, mmol/L | | | | | | | | | | | | | | | |
| Average total MET- | | | | | | | | | | | | | | | |
| minutes/week | | | | | | | | | | | | | | | |

Abbreviations: IQR, Interquartile Range; N, Number; SD, Standard Deviation.



### 16.4 Summary of categorical baseline characteristics

| Baseline | | rol group<br>n = ) | | tion group<br>n = ) | A CONTRACT OF THE SECOND | opulation<br>n = ) |
|---|---|---|---|---|---|---|
| characteristic | Number | Percentage | Number | Percentage | Number | Percentage |
| Sex | | | | | | |
| Men | | | | | | |
| Women | | | | | | |
| Missing | | | | | | |
| Ethnicity | | | | | | |
| [TBC] | | | | | | |
| [TBC] | | | | | | |
| [TBC] | | | | | | |
| Missing | | | | | | |
| Smoking status | | | | | | |
| Never smoker | | | | | | |
| Ex-smoker | | | | | | |
| Current smoker | | 2015 | | | | |
| Missing | | | | | | |
| Glycaemic Status | | | | | | |
| Normoglycaemia | | | | | | |
| Prediabetes | | | | | | |
| Diabetes | | | | | | termina and the day of |
| Diabetes remission | | | | | | |
| Missing | | | | | | |
| Hypertension status | | | | | | |
| No | | | | | | |
| Yes | | | | | | |
| Missing | | | | | | |
| Sleep apnoea status | | | | | | |
| No | | | | | | |
| Yes | | | | | | |
| Missing | | | | | | |
| Total number of medications | | | | | | |
| 0 | | | | | | |
| 1 | | | | 7.574557463 | | |



| Baseline | | ol group<br>n = ) | | tion group<br>n = ) | | opulation<br>n = ) |
|---|---|---|---|---|---|---|
| characteristic | Number | Percentage | Number | Percentage | Number | Percentage |
| 2 | 70 | | | | | |
| ≥3 | | | | | | |
| Missing | | | | | | |
| Number of diabetes medications | | | | | | |
| 0 | | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| ≥3 | | | | | | |
| Missing | | | | | | |
| Type of diabetes medication | | | | | | |
| SGLT-2 | | | | | | |
| Metformin | | | | | | |
| Sulphonylureas | | | | | | |
| Glitazones | | | | | | |
| Missing | | | | | | |
| Number of antihypertensive medications | | | | | | No Micro |
| 0 | | | | | | |
| 1 | | | | | | |
| 2 | | | | | | |
| ≥3 | | | | | | |
| Missing | | | | | | |
| CPAP use | | | | | | |
| No | | | | | | |
| Yes | | | | | | |
| Missing | | | | | | |
| Statin use | | | | | | |
| No | | | | | | |
| Yes | | | | | | |
| Missing | | | | | | |



# 16.5 Comparison of continuous baseline characteristics between those with and without primary outcome data

| Missi | ng prima<br>(r | ry out<br>1 = ) | come data | | Non-mis | | nary o<br>ı = ) | utcome da | ita | P-value <sup>a</sup> |
|---|---|---|---|---|---|---|---|---|---|---|
| N missing | Mean | SD | Median | QR | N missing | Mean | SD | Median | Į | |
| | N missing | Missing prima (r N missing Mean | Missing primary out (n = ) N missing Mean SD | Missing primary outcome data (n = ) N missing Mean SD Median | Mean SD Median | Mean SD Median IQR Nr | mg primary outcome data (n =) Mean SD Median IQR N missing Me Mean IQR N missing Me | mg primary outcome data (n =) Mean SD Median IQR N missing Me Mean IQR N missing Me | mg primary outcome data (n =) Mean SD Median IQR N missing Me Mean IQR N missing Me | ng primary outcome data (n = ) Mean SD Median IQR N missing Mean SD Median Mean SD Median IQR N missing Mean SD Median |



| | | | | | | | | | | | | reek | minutes/week |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | | MET- | total | Average total MET- |
| | Į<br>QR | lean SD Median IQR | SD | 12 | N missing Mean SD Median IQR N missing | IQR | Median | SD | Mean | N missing | | | |
| | | | n = ) | r) | | | | (n = ) | (r | | ristic | Baseline characteristic | Baseline |
| P-value | ta | g primary outcome data | nary o | sing prim | Non-missing | | Missing primary outcome data | ry out | ng prima | Missi | | | |

Abbreviations: IQR, Interquartile Range; N, Number; SD, Standard Deviation.

<sup>&</sup>lt;sup>a</sup> P-values were estimated using a t-test for normally distributed variables and a Mann-Whitney test for non-normally distributed variables.



### 16.6 Comparison of categorical baseline characteristics between those with and without primary outcome data

| Baseline<br>characteristic | outco | g primary<br>ome data<br>n = ) | outco | ing primary<br>me data<br>n = ) | P-value <sup>a</sup> |
|---|---|---|---|---|---|
| | Number | Percentage | Number | Percentage | |
| Sex | | | | | |
| Men | | | | | |
| Women | | | | | |
| Missing | | | | | |
| Ethnicity | | | | | |
| [TBC] | | | | | |
| [TBC] | | | | | |
| [TBC] | | | | | |
| Missing | | | | | |
| Smoking status | | | | | |
| Never smoker | | | | | |
| Ex-smoker | | | | | |
| Current smoker | | | | | |
| Missing | | | | | |
| Glycaemic Status | | | | | |
| Normoglycaemia | | | | | |
| Prediabetes | | | | | |
| Diabetes | | | | | |
| Diabetes remission | | | | | |
| Missing | | | | | |
| Hypertension status | | | | | |
| No | | | | | |
| Yes | | | | | |
| Missing | | | | | |
| Sleep apnoea status | | | | | |
| No | | | | | |
| Yes | | | | | |
| Missing | | | | | |
| Total number of medications | | | | | |
| 0 | | | | | |
| 1 | ECKNOWN | | | | |



| Baseline<br>characteristic | outco | g primary<br>ome data<br>n = ) | outco | ing primary<br>me data<br>1 = ) | P-value <sup>a</sup> |
|---|---|---|---|---|---|
| | Number | Percentage | Number | Percentage | |
| 2 | | | | | |
| ≥3 | | | | | |
| Missing | | | | | |
| Number of diabetes medications | | | | | |
| 0 | | | | | |
| 1 | | | | | |
| 2 | | | | | |
| ≥3 | | | | | |
| Missing | | | | | |
| Type of diabetes medication | | | | | |
| SGLT-2 | | | | | |
| Metformin | | | | | |
| Sulphonylureas | | | | | |
| Glitazones | | | | | |
| Missing | | | | | |
| Number of | | | | | |
| antihypertensive medications | | | | | |
| 0 | | | | | |
| 1 | | | | | |
| 2 | | | | | |
| ≥3 | | | | | |
| Missing | | | | | |
| CPAP use | | | | | |
| No | | | | | |
| Yes | | | | | |
| Missing | | | | | |
| Statin use | | | | | |
| No | | | | | |
| Yes | | | | | |
| Missing | | | | | |

<sup>&</sup>lt;sup>a</sup> P-values were estimated using a chi-squared test.

UNIVERSITY OF LEICESTER

### 16.7 Analysis of primary outcome

| Don: lation | | Control | | | Intervention | | between the two groups <sup>a</sup> | itterence<br>two groups <sup>a</sup> |
|---|---|---|---|---|---|---|---|---|
| N | N with | N with | % with | N with | N with | % with | OB (05% CI) | D value |
| d | data | outcome | outcome | data | outcome | outcome | OR (95% CI) P-value | P-value |
| Complete cases <sup>b</sup> | | | | | | | | |
| Intention-to-treat | | | | | | | | |
| Per protocol | | | | | | | | |
| Responder | | | | | | | | |

Abbreviations: Cl, Confidence Interval; OR, Odds Ratio.

<sup>&</sup>lt;sup>a</sup> Estimates are adjusted for the stratification variables: site and baseline body mass index (>45kg/m²; <45kg/m²).

<sup>&</sup>lt;sup>b</sup> Primary analysis

16.8 Analysis of secondary categorical anthropometric outcomes

| | | Control | | | Intervention | 3 | Adjusted difference between the two | fference<br>he two |
|---|---|---|---|---|---|---|---|---|
| | N with | N with | % with | N with | N with | % with | OR (95% CI) | P-value |
| Weight loss of ≥5% | | | | | | | | |
| 16 weeks | | | | | | | | |
| 32 weeks | | | | | | | | |
| 52 weeks | | | | | | | | |
| 104 weeks | | | | | | | | |
| Weight loss of ≥10% | | | | | | | | |
| 16 weeks | | | | | | | | |
| 32 weeks | | | | | | | | |
| 52 weeks | | | | | The second | INTO SERVICE | | |
| 104 weeks | | | | | | | | |
| Weight loss of ≥15% | | | | | | | | |
| 16 weeks | | | | | | | | |
| 32 weeks | | | | | | | | |
| 52 weeks <sup>b</sup> | | | | | | | | |
| 104 weeks | | | | | | | | |
| Maintenance of weight loss of ≥15% among those | | | | | | | | |



| | | | | | | | The second secon | |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | | 104 weeks |
| | | | | | | | | who lost ≥15% at 52 weeks |
| | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | outcome | outcome | data | outcome | outcome | data | |
| 7-VAILE | OK 195% C | | | | | | | |
| , | OB (05% CI) | % with | N with | N with | % with | N with | N with | |
| ps <sup>d</sup> | groups | | | | | | | Outcome |
| , | | | | | | | | |
| the two | between the two | ח | Intervention | | | Control | | |
| ifference | Adjusted difference | | | | | | | |

Abbreviations: Cl, Confidence Interval; OR, Odds Ratio.

<sup>b</sup> Primary analysis.

<sup>&</sup>lt;sup>a</sup> Estimates are adjusted for the stratification variables: site and baseline body mass index (>45kg/m²; <45kg/m²).



## 16.9 Analysis of secondary continuous anthropometric outcomes

| | B | Baseline | Fo | Follow-up | Change | Change from baseline | Difference in change from baseline | rom baseline |
|---|---|---|---|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention | Control | Intervention | Adjusted mean<br>difference (95% CI) <sup>a</sup> | P-value |
| Absolute weight (kg) at 16 weeks | 16 weeks | | | | | | | |
| Number | | | | | | | | |
| Mean | | | | | | | | |
| SD | | | | | | | , | ı |
| Median | | | | | | | | |
| Range | | | | | | | - | 1 |
| Interquartile range | | | | | | | | |
| Absolute weight (kg) at 32 weeks | 32 weeks | | | | | | | |
| Number | | | | | | | | |
| Mean | | | | | | | | |
| SD | | | | | | | | |
| Median | | | | | | | | 1 |
| Range | | | | | | | | |
| Interquartile range | | | | | | | 1 | 1 |
| Absolute weight (kg) at 52 weeks | 52 weeks | | | | | | | |
| Number | | | | | | | | |
| Mean | | | | | | | | |
| SD | | | | | | | • | _ |



| | В | Baseline | Fo | Follow-up | Change | Change from baseline | Difference in change from baseline | from baseline |
|---|---|---|---|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention | Control | Intervention | Adjusted mean<br>difference (95% CI) <sup>a</sup> | P-value |
| Median | | | | | | | | • |
| Range | | | | | | | 1 | 1 |
| Interquartile range | | | | | | | • | • |
| Absolute weight (kg) at 104 weeks | )4 weeks | | | | | | | |
| Number | | | | | | | | |
| Mean | | | | | | | | |
| SD | | | | | | | | |
| Median | | | | | | | 1 | 1 |
| Range | | | | | | | | |
| Interquartile range | | | | | | | • | 1 |
| Relative change in weight (%) at 16 weeks | (%) at 16 w | eeks | | | | | | |
| Number | | | | | | | | |
| Mean | • | | | | | | | |
| SD | 1 | • | ı | 1 | | | • | • |
| Median | | • | • | - | | | | • |
| Range | | 1 | • | | | | | |
| Interquartile range | 1 | • | | | | | | |
| Relative change in weight (%) at 32 weeks | (%) at 32 w | eeks | | | | | | |
| Number | | | Service of the service of the servic | Same and the second | | | | |
| Mean | 1 | • | • | | | | | |

| | В | Baseline | Fo | Follow-up | Change | Change from baseline | Difference in change from baseline | from ba |
|---|---|---|---|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention | Control | Intervention | Adjusted mean difference (95% CI) <sup>a</sup> | 1000 |
| SD | | | - | • | | | | • |
| Median | 1 | ı | • | 1 | | | 1 | |
| Range | 1 | | | | | | • | 1 |
| Interquartile range | 1 | ı | 1 | 1 | | | 1 | 1 |
| Relative change in weight (%) at 52 weeks | t (%) at 52 w | eeks | | | | | | |
| Number | | | | | | | | |
| Mean | • | | | • | | | | |
| SD | , | 1 | 1 | 1 | | | - | 1 |
| Median | • | ı | | - | | | | • |
| Range | 1 | 1 | 1 | 1 | | | 1 | |
| Interquartile range | • | | , | | | | • | • |
| Relative change in weight (%) at 104 weeks | t (%) at 104 | weeks | | | | | | |
| Number | | | | | | | | |
| Mean | ŧ | 1 | ı | ı | | | | |
| SD | | | • | • | | | | 1 |
| Median | 1 | 1 | 1 | 1 | | | • | 1 |
| Range | | | 1 | | | | | |
| Interquartile range | 1 | 1 | 1 | 1 | | | | 1 |
| Absolute BMI (kg/m²) at 52 weeks | 52 weeks | | | | | | | |
| Nimbor | | | | | | | | |



| SD Median Range Interquartile range Absolute waist circumference (cm) at 52 weeks Number Mean SD Median Range | Mean Control Intervention Control Intervention Control Median Median Intervention Control Range Interquartile range Absolute BMI (kg/m²) at 104 weeks Number Number |
|---|---|
| | Change from baseline Intervention |
| | Difference in change from baseline Adjusted mean difference (95% CI) <sup>a</sup> |



| | В. | Baseline | Fo | Follow-up | Change | Change from baseline | Difference in change from baseline | rom baseline |
|---|---|---|---|---|---|---|---|---|
| Outcome | Control | Control Intervention Control Intervention Contr | Control | Intervention | Control | Intervention | Adjusted mean<br>difference (95% CI) <sup>a</sup> | P-value |
| Number | | | | | | | | |
| Mean | | | | | | | | |
| SD | | | | | | | 1 | |
| Median | | | | | | | - | 1 |
| Range | | | | | | | | |
| Interquartile range | | | | | | | 1 | • |

Abbreviations: BMI, Body Mass Index; CI, Confidence Interval; OR, Odds Ratio.

<sup>&</sup>lt;sup>a</sup> Estimates are adjusted for the stratification variables: site and baseline body mass index (≥45kg/m²; <45kg/m²).



### **16.10** Summary of other categorical secondary outcomes

| Outcome | N (%) | at baseline | N (%) a | t follow-up |
|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention |
| King's College Obesity Staging Sy | stem at 52 | weeks | | |
| Normal health | | | | |
| At risk of disease | | | | |
| Established disease | | | | |
| Advanced disease | | | | |
| Missing | | | | |
| King's College Obesity Staging Sys | stem at 104 | l weeks | | |
| Normal health | | | | |
| At risk of disease | | | | |
| Established disease | | | | |
| Advanced disease | | | | |
| Missing | | | | |
| Patient health questionnaire-9 at | 52 weeks | | | |
| Minimal depression | | | | |
| Mild depression | | | | |
| Moderate depression | | | | |
| Moderately severe depression | | | | |
| Severe depression | | | | |
| Missing | | | | |
| Patient health questionnaire-9 at | 104 weeks | 100000000000000000000000000000000000000 | | |
| Minimal depression | | | | |
| Mild depression | | | | |
| Moderate depression | | | | |
| Moderately severe depression | | | | |
| Severe depression | | | | |
| Missing | | | | |
| Epworth sleepiness scale at 52 w | eeks | | | |
| No OSA | | | | |
| Possible OSA | | | | |
| Missing | | | | |
| Epworth sleepiness scale at 104 v | veeks | | | |
| No OSA | | | | |
| Possible OSA | | | | |
| Missing | | | | |
| Stop bang questionnaire at 52 we | eeks | | | |



N (%) at baseline N (%) at follow-up Outcome Control Intervention Control Intervention No OSA **Possible OSA Likely OSA** Missing Stop bang questionnaire at 104 weeks No OSA **Possible OSA** Likely OSA Missing On CPAP at 52 weeks No Yes Missing On CPAP at 104 weeks No Yes Missing Glycaemic Status at 52 weeks Normoglycaemia **Prediabetes Diabetes Diabetes remission** Missing Glycaemic Status at 104 weeks Normoglycaemia **Prediabetes Diabetes Diabetes remission** Missing Hypertension at 52 weeks No Yes Missing Hypertension at 104 weeks No Yes Missing

Referred to Tier 4 for bariatric surgery by 104 weeks



| Outcome | N (%) | at baseline | N (%) at follow-up | |
|---------|---------|--------------|--------------------|--------------|
| Outcome | Control | Intervention | Control | Intervention |
| No | | | | |
| Yes | | | | |
| Missing | | | | |

Abbreviations: CPAP, XX; N, Number; OSA, Obstructive Sleep Apnoea.

Trial:

STRIVE

SAP Version: 1.1 DRAFT Version Date: 01/08/2022



### 16.11 Summary of other secondary continuous outcomes

| 等 医克里斯氏征 多果 | В | aseline | Follow-up | | Change from ba | |
|---|---|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention | Control | Inter |
| EQ5D – Mobility at 52 wee | eks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| EQ5D - Mobility at 104 w | eeks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| EQ5D – Self-care at 52 we | eks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | The Market State | | E AMERICA | | | |
| EQ5D – Self-care at 104 w | eeks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | Shaai |
| Interquartile range | | | | | | |
| EQ5D – Usual activities at | 52 weeks | | | | STEEL STEEL | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |



| | В | aseline | Follow-up | | Change from ba | |
|---|---|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention | Control | Interv |
| Interquartile range | | | | | | |
| EQ5D – Usual activities at | 104 weeks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| EQ5D - Pain/discomfort a | t 52 weeks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | 9276 | | | |
| EQ5D - Pain/discomfort a | t 104 weeks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | <u> </u> | | | |
| EQ5D - Anxiety/depression | on at 52 weeks | The state of the s | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| EQ5D - Anxiety/depression | on at 104 week | KS. | | 200000000000000000000000000000000000000 | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | Le | |
| Range | | | | | | |
| Interquartile range | | | A STOCK STATE OF STAT | | | |
| EQ5D – VAS at 52 weeks | | | | | Rand Card Card | |


| | В | aseline | Fo | llow-up | Change | from ba |
|---|---|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention | Control | Interv |
| Number | | | | | | 35 FIRST VIEW (CO.) |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| EQ5D – VAS at 104 weeks | | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | distant a second |
| Range | | | | | Thymself ( | |
| Interquartile range | | | | | | |
| Impact of Weight on Quali | ty of Life-Lite a | at 52 weeks | | | CES BREAK | 10 2 0 |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | Jana Ball | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Impact of Weight on Quali | ty of Life-Lite a | at 104 weeks | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | TENSON DELISATION | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| <b>Patient Health Questionna</b> | ire-9 at 52 we | eks | | | | |
| Number | | | | | | |
| Mean | | | | | | N. Contraction |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | N. C. | | | | | |
| Patient Health Questionna | ire-9 at 104 w | eeks | Parallel Street Street Street Street | The second second | | |
| Number | | | | | | |



| <b>10世界的关系的</b> | В | aseline | Fo | llow-up | Change | ange from ba |
|---|---|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention | Control | Inter |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Epworth Sleepiness Scale at ! | 52 weeks | | VI STATE OF | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Epworth Sleepiness Scale at : | 104 weeks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Stop Bang score at 52 weeks | | | | | | |
| Number | | | | Lieuwa na | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Stop Bang score at 104 week | (S | | | | | |
| Number | | | | | | |
| Mean | | | | | 1 1 2/1 | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | - West F | |
| CPAP compliance – Average | hours per o | lay at 52 weeks | | | | |
| Number | | TO DESCRIPTION | | Line of the | | |
| Mean | | | | | | |

Trial: SAP Version: 1.1 DRAFT

**STRIVE** Version Date: 01/08/2022



| | В | aseline | Fo | llow-up | Change | from ba |
|---|---|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention | Control | Inter |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | Mary 1 | | | on state |
| CPAP compliance – Averag | ge hours per da | y at 104 weeks | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| HbA1c (mmol/mol) at 52 v | veeks | | | | all moderns | (Valle) |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| HbA1c (mmol/mol) at 104 | weeks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | Apple 18 San Carlo | |
| Interquartile range | | | | | | |
| HbA1c (%) at 52 weeks | | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| HbA1c (%) at 104 weeks | | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | STRUM. |



| | В | aseline | Fo | llow-up | Change | e from ba |
|---|---|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention | Control | Inter |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Total number of agents for | r diabetes at 5 | 2 weeks | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Total number of agents fo | r diabetes at 1 | 04 weeks | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Albumin-creatinine ratio ( | mg/mmol) at | 52 weeks <sup>a</sup> | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Albumin-creatinine ratio ( | mg/mmol) at | 104 weeks <sup>a</sup> | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | 10.11-1 | |
| Systolic blood pressure (n | nmHg) at 52 w | eeks | | Karacara Pos | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |

Trial:



| | В | aseline | Fo | llow-up | Change | from ba |
|---|---|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention | Control | Interv |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Systolic blood pressure (m | mHg) at 104 w | reeks | | | | |
| Number | | | | | The state of the | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Diastolic blood pressure (n | nmHg) at 52 w | eeks | | | | ON SAC SA |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Diastolic blood pressure (m | nmHg) at 104 v | weeks | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | (Section ) | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Total number of agents for | hypertension | at 52 weeks | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Total number of agents for | hypertension | at 104 weeks | No. | | Control of the last | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | 4 | | |
| Median | | | | | | |
| Range | | | | | | |



| | В | aseline | Fo | llow-up | Change | from b |
|---|---|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention | Control | Inter |
| Interquartile range | | | | | | _ |
| LDL cholesterol (mmol/L) at | 52 weeks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| LDL cholesterol (mmol/L) at | 104 weeks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| HDL cholesterol (mmol/L) at | 52 weeks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| HDL cholesterol (mmol/L) a | t 104 weeks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | i i i i | |
| Total cholesterol (mmol/L) | at 52 weeks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Total cholesterol (mmol/L) | at 104 wook | 6 | | | | - |



| | В | aseline | Fo | llow-up | Change | from b |
|---|---|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention | Control | Inter |
| Number | | | | | | |
| Mean | | | | | - | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | - | |
| Triglycerides (mmol/L) at | 52 weeks | | | | | |
| Number | | | | | - 1.1 | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Triglycerides (mmol/L) at | 104 weeks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | 7 | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Total number of agents for | or dyslipidaemi | ia at 52 weeks | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | A CHARLES | | MINISTER STATE | |
| Total number of agents for | or dyslipidaem | ia at 104 weeks | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| <b>Treatment Satisfaction Q</b> | uestionnaire fo | or Medication (T | SQM) at 52 | weeks | | |
| Number | | | | | | |



| | В | aseline | Fo | Follow-up Cha | | nge from ba |
|---|---|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention | Control | Interv |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Treatment Satisfaction Qu | estionnaire fo | r Medication (TS | QM) at 10 | 4 weeks | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | <u> </u> |
| Range | | | | | | |
| Interquartile range | | | | | | - |
| Total MET-minutes/week a | t 52 weeks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | <del></del> | | | | |
| Interquartile range | | | | | | dia sise |
| Total MET-minutes/week a | t 104 weeks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |

Abbreviations: VAS, Visual Analogue Scale.

<sup>&</sup>lt;sup>a</sup> Only defined for participants with diabetes, prediabetes, or hypertension.

Trial:

STRIVE

SAP Version: 1.1 DRAFT Version Date: 01/08/2022



### 16.12 Summary of categorical safety outcomes

| Outcome | N (%) | at baseline | N (%) at follow-up | |
|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention |
| Gastrointestinal symptoms within | n 52 weeks | | | |
| No | | | | |
| Yes | | | | |
| Missing | | | | |
| Gastrointestinal symptoms within | 104 week | S | | |
| No | | | | |
| Yes | | | | |
| Missing | | | | |



## 16.13 Summary of continuous safety outcomes

| | В | aseline | Fo | llow-up | Change | |
|---|---|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention | Control | Inte |
| Overall hypoglycaemia rate – | ADA defini | tion at 52 week | | | | |
| Number | | | | | | THE STREET |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Overall hypoglycaemia rate – | ADA defin | ition at 104 wee | ks | | | |
| Number | | | | | | |
| Mean | | | 200 | | | |
| SD | | | | | | 100 H (6-18 |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Overall hypoglycaemia rate – | Novo Nor | disk definition a | t 52 weeks | | | 28181-221- |
| Number | | | | | | |
| Mean | | | - | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Overall hypoglycaemia rate - | - Novo No | rdisk definition a | it 104 week | (S | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Overall adverse event rate a | t 52 weeks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | to Simon School | | | | X-1 |
| Range | | | | | | |
| Interquartile range | | | | | | |



| | В | aseline | | | | ge from b |
|---|---|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention | Control | Inte |
| Overall adverse event rate | e at 104 weeks | | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | The state of the s | | n comenia | | |
| Interquartile range | | | | | | |
| Overall serious adverse e | vent rate at 52 | weeks | | | | |
| Number | | | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | ENERGY STATE | | |
| Overall serious adverse e | vent rate at 10 | 4 weeks | | | | |
| Number | Vene rate at 20 | THE STATE OF THE S | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Overall severe hypoglyca | omia event rat | e at 52 weeks | | | | |
| Number | elilla evelit lat | e at 52 WCCR3 | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Overall severe hypoglyca | omia event rat | e at 104 weeks | | | | |
| Number | eilla event rat | e at 104 weeks | | | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | to be the first on the second | |
| Range | | 2 医自由 中国 自由 1000 1000 1000 1000 1000 1000 1000 1 | | | | |
| Interquartile range | unto) at E2 was | also | | | | 56919 |
| Heart rate (beats per mir<br>Number | iutej at 52 wee | CA: | | | | T |

Trial: STRIVE


SAP Version: 1.1 DRAFT



| | В | aseline | Follow-up | | Change from | |
|---|---|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention | Control | Interv |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |
| Heart rate (beats per min | ute) at 104 wee | eks | | | | |
| Number | | | | Approximation | | |
| Mean | | | | | | |
| SD | | | | | | |
| Median | | | | | | |
| Range | | | | | | |
| Interquartile range | | | | | | |



### 16.14 Summary of categorical compliance outcomes

| | N (%) | at baseline | N (%) a | t follow-up |
|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention |
| Attended at least 70% of schedu | uled Tier 3 ap | pointments at | 52 weeks | |
| No | | | | |
| Yes | | | | |
| Missing | | | | |
| Attended at least 70% of sched | uled Tier 3 ap | pointments at | 104 weeks | |
| No | | | | |
| Yes | | | | |
| Missing | | | | |
| Stopped treatment with LIRA 3 | mg due to ad | verse effects a | t 52 weeks | |
| No | | | | |
| Yes | | | | |
| Missing | | | | |
| Stopped treatment with LIRA 3 | mg due to ad | lverse effects a | t 104 weeks | |
| No | | | | |
| Yes | | | | |
| Missing | | | | |
| Compliant with LIRA 3mg treat | ment at 52 w | reeks | | |
| No | | | | |
| Yes | | | | |
| Missing | | | | |
| Compliant with LIRA 3mg treat | ment at 104 | weeks | | |
| No | | | | |
| Yes | | | | |
| Missing | | | | |
| Stopped LIRA 3mg treatment a | t 16 weeks | | | |
| No | | | | |
| Yes | | | | |
| Missing | | | | |
| Stopped LIRA 3mg treatment a | t 32 weeks | | | |
| No | | | | |
| Yes | | | | |
| Missing | | | | |
| Stopped LIRA 3mg treatment a | t 52 weeks | | | |
| No | | | | |
| Yes | | | | |



| | N (%) | at baseline | N (%) a | t follow-up |
|---|---|---|---|---|
| Outcome | Control | Intervention | Control | Intervention |
| Missing | | | | |
| Completed 52 weeks of the | Tier 3 programm | e despite stopp | ing LIRA 3n | ng at 16 weeks |
| No | | | | |
| Yes | | | | |
| Missing | | | | |
| Completed 52 weeks of the | Tier 3 programn | ne despite stopp | ing LIRA 3n | ng at 32 weeks |
| No | | | | |
| Yes | | | | |
| Missing | | | | |
| Started on anti-obesity drug | gs at 52 weeks | | | |
| No | | | | |
| Yes | | | | |
| Missing | | | | |
| Started on anti-obesity drug | gs at 104 weeks | | | |
| No | | | | |
| Yes | | | | |
| Missing | | | | |



# 16.15 Summary of Adverse events by MEDRA and expected adverse event terms

Incidence rate (per person year) of each System Organ Class of AEs by treatment and Overall

| Overall | | | | | | | Name and Address of the Owner, where the Owner, which is the Owner, which is the Owner, where the Owner, which is the Owner, |
|---|---|---|---|---|---|---|---|
| | Sta | ndard | Lira | glutide | Ove | rall | |
| System Organ Class | N | Incidenc | N | Incidence | N | Incidenc | Incidence |
| | | е | | | | е | Rate Ratio |
| Blood and lymphatic system | | | | | | | |
| disorders | | | | | | | |
| Cardiac disorders | | | | | | | |
| Congenital, familial and genetic disorders | | | | | | | |
| Ear and labyrinth disorders | | | | | | | |
| Endocrine disorders | | | | | | | |
| •••• | | | | | | | |

### Proportion of patients with at least one AE, by SOC type, treatment arm and overall

| | Stand | lard | Liraglu | ıtide | Overall | |
|---|---|---|---|---|---|---|
| System Organ Class | N | % | N | % | N | % |
| Blood and lymphatic system disorders | | | | | | |
| Cardiac disorders | | | | | | |
| Congenital, familial and genetic disorders | | | | | | |
| Ear and labyrinth disorders | | | | | | |
| Endocrine disorders | | | | · | | |
| •••• | | | | | | |



### Incidence rate (per person year) of each Expected AE Type by treatment and Overall

| Expected AE Type | Star<br>N | ndard<br>Incidence | Liraglu<br>N | tide<br>Incidence | Over<br>N | all<br>Incidence | Incidence<br>Rate<br>Ratio |
|---|---|---|---|---|---|---|---|
| N/A | | | | | | | |
| Anaphylactic reaction | | | | | | | |
| Hypoglycaemia | | | | | | | |
| Dehydration | | | | | | | |
| Dizziness | | | | | | | |
| Nausea | | | | | | | |

# Proportion of patients with at least one expected AE, by AE type, treatment arm and overall

| over un | Standar | d | Liraglut | ide | Overal | |
|-----------------------|---------|---|----------|-----|--------|---|
| Expected AE Type | | % | N | % | N | % |
| N/A | | | | | | |
| Anaphylactic reaction | | | | | | |
| Hypoglycaemia | | | | | | |
| Dehydration | | | | | | |
| Dizziness | | | | | | |
| Nausea | | | | | | |
| •••• | | | | | | |



### Proportion of individuals with at least one AE of given Severity by treatment and overall

| | Standa | rd | Liraglut | ide | Overal | |
|----------|--------|----|----------|-----|--------|---|
| Severity | N | % | N | % | N | % |
| Mild | | | | | | |
| Moderate | | | | | | |
| Severe | | | | | | |
| Fatal | | | | | | |

## Proportion of individuals with at least one AE of given Likelihood Related by treatment and overall

| | Standa | rd | Liraglut | ide | Overal | |
|-----------------------|--------|----|----------|-----|--------|---|
| Likelihood<br>Related | N | % | N | % | N | % |
| Not Related | | | | | | |
| Unlikely | | | | | | |
| Possible | | | | | | |
| Probable | | | | | | |
| Definite | | | | | | |



# Incidence rate (per person year) of each System Organ Class of SAEs by treatment and Overall

| HICKORY CONTRACTOR STATE | Act Lan | and the state of t | | | | | |
|---|---|---|---|---|---|---|---|
| | Stan | Standard | Lirag | Liraglutide | Overall | rall | |
| System Organ Class | Z | Incidence | z | Incidence N Incidence | Z | N Incidence | Incidence Rate |
| | | | | | | | Ratio |
| Blood and lymphatic | 100 | | | | | | |
| system disorders | | | | | | | |
| Cardiac disorders | | | | | | | |
| Congenital, familial | | | | | | | |
| and genetic disorders | | | | | | | |
| Ear and labyrinth | | | | | | | |
| disorders | | | | | | | |
| <b>Endocrine disorders</b> | | | | | | | |

UNIVERSITY OF LEICESTER

Trial: STRIVE
SAP Version: 1.1 DRAFT

# Proportion of patients with at least one SAE, by SOC type, treatment arm and overall

| • | <b>Endocrine disorders</b> | disorders | Ear and labyrinth | and genetic disorders | Congenital, familial | Cardiac disorders | system disorders | Blood and lymphatic | System Organ Class | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | N % | Standard |
| | | | | | | | | | N % | Liraglutide |
| | | | | | | | | | N % | Overall |



# Incidence rate (per person year) of each Expected SAE Type by treatment and Overall

| | 11. | | | | | , | | |
|---|---|---|---|---|---|---|---|---|
| | Star | Standard | Lira | Liraglutide | Ove | Overall | | |
| Expected AE Type | Z | N Incidence N Incidence | z | | z | N Incidence Incidence | Incidence | |
| | | | | | | | Rate Ratio | |
| N/A | | | | | | | | 10 |
| Anaphylactic reaction | | | | | | | | |
| Hypoglycaemia | | | | | | | | 1 |
| Dehydration | | | | | | | | |
| Dizziness | | | | | | | | L |
| Nausea | | | | | | | | 1 |
| | | | | | | | | 1 |

# Proportion of patients with at least one expected SAE, by AE type, treatment arm and overall

| | Standard | ard | Liraglutide | utide | Overall | all |
|---|---|---|---|---|---|---|
| Expected AE Type | Z | % | Z | % | Z | % |
| N/A | | | | | | |
| Anaphylactic reaction | | | | | | |
| Hypoglycaemia | | | | | | |
| Dehydration | | | | | | |
| Dizziness | | | | | | |
| Nausea | | | | | | |
| | - | | | | | |

UNIVERSITY OF LEICESTER

